# Statistical Analysis Plan



| Sponsor: | KemPharm, Inc. |
|---|---|
| Protocol Title: | A Multicenter, Dose-Optimized, Open-Label Safety Study with KP415 in Children with Attention-Deficit/Hyperactivity Disorder |
| Protocol Number: | KP415.S01 |
| Premier Research PCN: | KEMP7419 |
| Document Version: | Final 1.0 |
| Document Date: | 01-Aug-2018 |

# **Approvals**

| Role | Signatures | Date (dd-Mmm-yyyy) |
|---|---|---|
| | Print Name: Adrienne Kuxhausen | |
| | Sign Name: | |
| Lead | | |
| Biostatistician | DocuSigned by: Figure Rushmusen | |
| | Signer Name: Adrienne Kuxhausen Signing Reason: I am the author of this document Signing Time: 01-Aug-2018 15:43:42 EDT | |
| | Print Name: Valeric Smith | |
| | Sign Name: | |
| Senior Reviewer | DocuSigned by: | |
| | Valerie Smith | |
| | Signer Name: Valerie Smith Signing Reason: I approve this document Signing Time: 01-Aug-2018 16:29:22 EDT | |
| | Print Name: Rene Braeckman | |
| | Sign Name: | |
| KemPharm, Inc. Representative | DocuSigned by: | |
| Representative | Pene Brackman | |
| | Signer Name: Rene Braeckman Signing Reason: I approve this document Signing Time: 02-Aug-2018 09:52:05 EDT | |





# **Document History**

Not applicable.





## **Table of Contents**

| Approvals | . 1 |
|-------------------------------------------------------|-----|
| Document History | . 2 |
| Table of Contents | . 3 |
| List of Tables | . 4 |
| List of Figures | . 5 |
| 1. Overview | . 6 |
| 2. Study Objectives and Endpoints | . 6 |
| 2.1. Study Objectives | . 6 |
| 2.1.1. Primary Objective | . 6 |
| 2.1.2. Secondary Objectives | . 6 |
| 2.2. Study Endpoints | . 6 |
| 2.2.1. Safety Endpoints | . 7 |
| 2.2.2. Efficacy Endpoints | . 7 |
| 2.2.3. Other Endpoint | . 7 |
| 3. Overall Study Design and Plan | . 8 |
| 3.1. Overall Design | . 8 |
| 3.2. Sample Size and Power | . 8 |
| 3.3. Study Population | . 8 |
| 3.4. Treatments Administered | . 8 |
| 3.5. Method of Assigning Subjects to Treatment Groups | . 8 |
| 3.6. Blinding and Unblinding | |
| 3.7. Schedule of Events | . 8 |
| 4. Statistical Analysis and Reporting | 17 |
| 4.1. Introduction | 17 |
| 4.2. Interim Analysis and Data Monitoring | 18 |
| 5. Analysis Populations | 18 |
| 6. General Issues for Statistical Analysis | 19 |
| 6.1. Statistical Definitions and Algorithms | 19 |
| 6.1.1. Baseline | 19 |
| 6.1.2. Adjustments for Covariates | 19 |
| 6.1.3. Multiple Comparisons | 19 |
| 6.1.4. Handling of Dropouts or Missing Data | 19 |
| 6.1.5. Analysis Visit Windows | 20 |
| 6.1.6. Pooling of Sites | 20 |
| 6.1.7. Derived Variables | 20 |
| 6.1.8. Data Adjustments/Handling/Conventions | 21 |
| AD-ST-33.05 Effective date: 22-Jan-2018 | |





| 7. | Stı | udy Subjects and Demographics | 22 |
|---|---|---|---|
| | 7.1. | Disposition of Subjects and Withdrawals | 22 |
| | 7.2. | Protocol Violations and Deviations | 23 |
| | 7.3. | Demographics and Other Baseline Characteristics | 23 |
| | 7.4. | Exposure and Compliance | 23 |
| 8. | Ef | ficacy Analysis | 24 |
| | 8.1. | Secondary Efficacy Analysis | 24 |
| 9. | Sa | fety and Tolerability Analysis | 25 |
| | 9.1. | Adverse Events | 25 |
| | 9.1.1. | Adverse Events Leading to Withdrawal | 26 |
| | 9.1.2. | Deaths and Serious Adverse Events | 26 |
| | 9.1.3. | Other Significant Adverse Events | 26 |
| | 9.2. | Clinical Laboratory Evaluations | 27 |
| | 9.3. | Vital Signs | 28 |
| | 9.4. | Electrocardiograms | 28 |
| | 9.5. | Further Safety Evaluations | 28 |
| | 9.6. | Concomitant Medication. | 28 |
| 10. | Ch | nanges from Planned Analysis | 29 |
| 11. | Ot | her Planned Analysis | 29 |
| 12. | Re | ferences | 30 |
| 13. | Ta | bles, Listings, and Figures | 30 |
| | 13.1. | Planned Table Descriptions | 30 |
| | 13.2. | Efficacy Data | 31 |
| | 13.3. | Safety Data | 33 |
| | 13.4. | Other Data Summary Tables | 36 |
| | 13.5. | Planned Listing Descriptions | 36 |
| | 13.6. | Planned Figure Descriptions | 38 |
| | 13.7. | Standard Layout for all Tables, Listings, and Figures | 39 |
| | 13.8. | Planned Table Shells | 41 |
| | 13.9. | Planned Listing Shells | 88 |
| | 13.10. | Planned Figure Shells | 113 |
| Ap | pendix | 1: Premier Research Library of Abbreviations | 114 |
| Li | st of T | <b>Sables</b> | |
| | | chedule of Events (Screening [all subjects] and Dose Optimization Phase [ne | w |





| Table 2: Schedule of Events (Treatment Phase [First 6 Months; All Subjects]) | . 13 |
|---|---|
| Table 3: Schedule of Events (Treatment Phase [Second 6 Months], and Early Termination and Follow-Up Visits [All Subjects]) | |
| Table 4: Demographic Data Summary Tables and Figures | . 31 |
| Table 5: Efficacy Data | . 31 |
| Table 6: Safety Data. | . 33 |
| Table 7: Planned Listings. | . 36 |
| List of Figures | |
| Figure 1: Standardized Layout | . 40 |





#### 1. Overview

This statistical analysis plan (SAP) describes the planned analysis and reporting for KemPharm, Inc. protocol number KP415.S01 (A Multicenter, Dose-Optimized, Open-Label Safety Study with KP415 in Children with Attention-Deficit/Hyperactivity Disorder), dated 26-Apr-2018, Amendment #2. Reference materials for this statistical plan include the protocol and the accompanying sample data collection documents. Operational aspects related to collection and timing of planned clinical assessments are not repeated in this SAP unless relevant to the planned analysis.

The structure and content of this SAP provides sufficient detail to meet the requirements identified by the Food and Drug Administration (FDA), European Medicines Agency (EMA), and International Conference on Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use: Guidance on Statistical Principles in Clinical Trials<sup>1</sup>. All work planned and reported for this SAP will follow internationally accepted guidelines, published by the American Statistical Association<sup>2</sup> and the Royal Statistical Society<sup>3</sup>, for statistical practice.

The planned analyses identified in this SAP may be included in clinical study reports (CSRs), regulatory submissions, or future manuscripts. Also, post-hoc exploratory analyses not necessarily identified in this SAP may be performed to further examine study data. Any post-hoc or unplanned, exploratory analysis performed will be clearly identified as such in the final CSR.

The statistical plan described hereafter is an *a priori* plan. It will be submitted to file prior to any unblinded inferential or descriptive analysis of data pertaining to KemPharm, Inc.'s study KP415.S01.

#### 2. Study Objectives and Endpoints

#### 2.1. Study Objectives

#### 2.1.1. Primary Objective

The primary objective is to determine the safety and tolerability of KP415 in treating children with attention-deficit hyperactivity disorder (ADHD).

#### 2.1.2. Secondary Objectives

The secondary objectives are to determine the efficacy and changes in sleep behavior during KP415 treatment in children with ADHD.

#### 2.2. Study Endpoints

This study is primarily an open-label safety study in the target patient population after approximately 12 months of daily oral doses of KP415 capsules, or after a shorter duration if the study is stopped at an interim analysis. Therefore, the primary endpoint is safety.



## 2.2.1. Safety Endpoints

The safety endpoints of this study include the following for all subjects:

- The occurrence of treatment-emergent adverse events (TEAEs) will be assessed starting following the first dose of study drug, and ending with the Follow-Up Visit or Early Termination Visit.
- Physical examinations will be performed at the first visit (at Screening, before the first dose of study drug), after approximately 6 months of treatment (Visit 11), and at the end of the Treatment Phase (Visit 17, End of Treatment [EOT]) or at Early Termination.
- Clinical laboratory tests will be performed at the first visit (at Screening, before the first dose of study drug), after approximately 6 months of treatment (Visit 11), and at the end of the Treatment Phase (Visit 17, EOT) or at Early Termination.
- Electrocardiogram (ECG) parameters will be collected at the first visit (at Screening, before the first dose of study drug), after approximately 6 months of treatment (Visit 11), and at the end of the Treatment Phase (Visit 17, EOT) or at Early Termination.
- Vital signs, height, weight, and body mass index (BMI) will be collected at each study visit.
- The Columbia-Suicide Severity Rating Scale (C-SSRS) will be performed at each study visit.

#### 2.2.2. Efficacy Endpoints

The efficacy endpoints of this study include the following:

- During the Dose Optimization Phase (new subjects only):
  - Clinical Global Impressions—Severity (CGI-S) will be assessed at each visit
    (Screening to Visit 5). Attention-Deficit Hyperactivity Disorder Rating Scale 5
    (ADHD-RS-5) will be administered at Visits 2 through Visit 5. Clinical Global
    Impressions—Improvement (CGI-I) will be assessed at Visits 3, 4, and 5 (since
    CGI-I is an ADHD improvement assessment, it will not be assessed at Screening
    and at Visit 2).
- During the Treatment Phase (all subjects):
  - o ADHD-RS-5 and CGI-S will be assessed at each visit (Visit 5 to Visit 17, EOT).

#### 2.2.3. Other Endpoint

The modified, abbreviated Children's Sleep Habits Questionnaire (CSHQ) will be used to assess the sleep behavior in the Dose Optimization Phase for new subjects (Visit 2) and in the Treatment Phase for all subjects (Visit 5 to Visit 17). The baseline will be measured before the first dose of study drug, at Visit 2 for new subjects and at Visit 5 for roll-over subjects.



## 3. Overall Study Design and Plan

## 3.1. Overall Design

## 3.2. Sample Size and Power

No formal sample size calculations were conducted. It was determined that approximately 200 subjects are adequate to satisfy the primary objective of the study, which is to determine the safety and tolerability of KP415 in treating children with ADHD for at least 6 months. Assuming a maximum dropout rate of 20% over 6 months, approximately 250 subjects will be enrolled. Subjects will be rolled over from Study KP415.E01 and to reach the targeted number of subjects, new subjects will be enrolled as well. Subjects who fail Screening and new subjects who terminate early during the Dose Optimization Phase may be replaced. Subjects who terminate early in the Treatment Phase will not be replaced.

#### 3.3. Study Population

The study population includes subjects rolled over from Study KP415.E01 (aged 6 to 13) or new subjects (aged 6 to 12) with ADHD who meet the inclusion/exclusion criteria listed in the protocol.

#### 3.4. Treatments Administered

All subjects will be administered 1 unblinded KP415 capsule once daily in the Treatment Phase. The dose of KP415 will be determined by the optimal dose of KP415 identified at the end of the Dose Optimization Phase, either 20, 30, or 40 mg/day KP415.

## 3.5. Method of Assigning Subjects to Treatment Groups

**Dose Optimization Phase (new subjects only):** All eligible subjects will start on a dose of 30 mg/day open-label KP415 and the KP415 dose will be titrated to either 20, 30 or 40 mg/day based on tolerability and best individual dose-response in the opinion of the Investigator.

**Treatment Phase (all subjects):** Roll-over subjects from Study KP415.E01, and new subjects who completed the Dose Optimization Phase (and passed the eligibility criteria for the Treatment Phase will be enrolled at Visit 5 (start of the Treatment Phase) for treatment with the optimized dose of KP415 capsules. During the Treatment Phase, based on individual tolerability and dose response, the daily dose of KP415 may be changed to any of the allowed dose levels (20, 30, or 40 mg/day) at the Investigator's discretion.

### 3.6. Blinding and Unblinding

This is an open-label study. Study treatments will not be blinded.

#### 3.7. Schedule of Events

A detailed schedule of events for the study is provided in Table 1 (Screening [all subjects] and Dose Optimization Phase [new subjects only]), Table 2 (Treatment Phase, first 6 months [all subjects]), and Table 3 (Treatment Phase, second 6 months; Early Termination; and Follow-up





Visits [all subjects]).





# Table 1: Schedule of Events (Screening [all subjects] and Dose Optimization Phase [new subjects only])

| ASSESSMENTS | NEW<br>SCREENING | PHASE <sup>22</sup><br>ROLLOVER | D | OPEN-LABEL<br>DOSE OPTIMIZATION PHASE <sup>21, 22</sup><br>(NEW SUBJECTS ONLY) | | | | |
|---|---|---|---|---|---|---|---|---|
| Study Day | -30 to | -30 to | 0 | 1-6<br>(±3<br>Days) | 7<br>(±3<br>Days) | 8-13<br>(±3<br>Days) | 14<br>(±3<br>Days) | 15-20<br>(±3<br>Days) |
| Visit Number | 1A | $1B^{24}$ | 2 | | 3 | | 4 | |
| Parental Permission/Written or Verbal<br>Assent | X | X | | | | | | |
| ADHD Diagnosis and Confirmation <sup>1</sup> | X | | | | | | | |
| Capsule Swallowing Test <sup>2</sup> | X | | | | | | | |
| Inclusion/Exclusion | X | X | X | | X | | X | |
| Demographics | X | X | | | | | | |
| Medical History <sup>3</sup> | X X | | X | | | | | |
| Physical Examination | X X | | | | | | | |
| Body Weight, Height, BMI <sup>4</sup> | X | X | | | | | | |
| Vital Signs <sup>5</sup> | X | X | X | | X | | X | |
| 12-Lead ECG <sup>6</sup> | X | X | | | | | | |
| Chemistry/Hematology/Urinalysis (under fasting conditions) | X | X | | | | | | |
| Urine Alcohol/Drugs of Abuse Screen <sup>7</sup> | X | X | | | | | | |
| Urine MPH Screen <sup>8</sup> | X | | X | | | | | |
| Pregnancy Test <sup>9</sup><br>C-SSRS <sup>10</sup> | X | X | X | | | | | |
| C-SSRS 10 | X | X | X | | X | | X | |
| Washout ADHD Meds 11 | | | X | | | | | |
| Open-Label KP415 Dosing <sup>12</sup> | | | | X | X | X | X | X |
| Drug Accountability & Compliance | | | | | X | | X | |
| Assessment 13 | | | 37 | | 37 | | 37 | |
| ADHD-RS-5 <sup>14</sup> | 37 | | X | | X | | X | |
| MINI-KID 15 | X | | 37 | | 37 | | 37 | |
| CGI-S <sup>16</sup> | X | | X | | X | | X | |
| CGI-I 17 | | | 37 | | X | | X | |
| CSHQ <sup>18</sup> | - | | X | 37 | 37 | 37 | 37 | 37 |
| Adverse Events 19 | 37 | | 37 | X | X | X | X | X |
| Concomitant Medications <sup>20</sup> | X | | X | | X | | X | |

BMI = Body Mass Index; ECG = Electrocardiogram; MPH = methylphenidate; see footnotes for other abbreviations.

- 1. ADHD Diagnosis based on the Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD (combined, inattentive, or hyperactive/impulsive presentation) and confirmed by the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
- 2. Capsule Swallowing Test: Subjects must be able to comply with one of the following:

Statistical Analysis Plan, Sponsor KemPharm, Inc. Protocol Number KP415.S01 PCN Number KEMP7419



- a) Subjects will take a size 3 capsule with up to 240 mL of water at Screening. The capsule may not contain any active drug substance. Subjects must be able to easily swallow the size 3 capsule to be eligible for further study participation. This is not required for subjects who have previously participated in the KP415.E01 study.
- b) If subjects are unable to demonstrate that they can swallow size 3 capsules, they must agree to take the capsule contents sprinkled over a small amount of applesauce or added to a small amount of water during the study.
- Any of the methods of administration may be used on any day of the study, but if subjects plan to take study drug as the whole capsule, subjects will need to have demonstrated that they are able to swallow size 3 capsules at Screening or any time during the study (or have been previously participated in Study KP415.E01).
- 3. Medical History: A complete medical history including chronic conditions, relevant surgical procedures (with start date), history of drug and alcohol use. As part of Medical History for Visit 1B (and with more details captured in the database), record treatment with study drug in Study KP415.E01 with regards to dose, duration, date of last dose (Visit 6 in Study KP415.E01), last visit in Study KP415.E01 (Visit 7 in Study KP415.E01), etc.
- 4. Height will be recorded in centimeters (cm) with the subject's shoes removed. Body weight will be measured in kilograms (kg); subjects will remain in their normal clothing with shoes and jacket (and/or outer clothing) removed.
- 5. Vital sign measurements will be obtained after the subject has been seated for at least 3 minutes. Vital signs will include sitting blood pressure (systolic and diastolic measurements), pulse rate (beats per minute), respiratory rate (breaths per minute), and oral temperature. Vital signs will be collected once at each visit.
- 6. Electrocardiogram (ECG): A 12-lead ECG will be obtained after the subject has been in the supine position for at least 3 minutes. Abnormal ECGs may be repeated for confirmation in which case only the repeated ECG will be recorded. The QT interval corrected for heart rate will be calculated with Fridericia's formula (QTcF). For roll-over subjects, if the Screening Visit (Visit 1B) occurs on the same day as the Follow-Up Visit (Visit 7) of Study KP415.E01, one ECG will be obtained to be used in both studies. If Visit 1B occurs later, after Visit 7 in E01, a new ECG will be obtained at Visit 1B as baseline for the current study.
- 7. Urine Screen for Alcohol and Drugs of Abuse: Urine samples will be tested for alcohol, and drugs of abuse (amphetamines, methamphetamines, benzodiazepines, barbiturates, cannabinoids, cocaine, opioids including oxycodone) at Screening (Visit 1A or 1B). If the urine test is positive for any of the analytes at Screening, the subject will be excluded from study participation, with the exception of the following: Depending on a subject's current ADHD medication at Screening, the urine screen at Screening may test positive for ADHD medications such as amphetamines and methamphetamines. All ADHD medications must be washed out by Visit 2 for new subjects and Visit 5 for roll-over subjects.
- 8. Urine Screen for Methylphenidate (MPH): For new subjects, urine samples will be tested for MPH at Screening (Visit 1A) and Visit 2. A urine dipstick (eg, NarcoCheck®) will be used to screen for the presence of MPH in the urine. If a subject's current ADHD medication at Screening contains MPH, the urine screen at Screening (Visit 1A, new subjects) may test positive for MPH. All ADHD medications must be washed out by Visit 2 for new subjects and Visit 5 for roll-over subjects (MPH urine screen must test negative).
- 9. Pregnancy Test: performed for female subjects of childbearing potential. A serum β-hCG pregnancy test will be performed at Screening. A urine pregnancy test will be performed at Visit 2. A positive pregnancy test at Screening or before the last dose of study drug will exclude a subject from further participation in the study.
- 10. Columbia-Suicide Severity Rating Scale (C-SSRS): The "Children's Baseline/Screening" version will be assessed at Screening, and the "Children's Since Last Visit" version will be assessed at all other visits. Subjects who have, in the opinion of the Investigator, clinically significant suicidal ideation/behavior, based on history of attempted suicide and the C-SSRS assessment at Screening or at any time before the last dose of study drug, will be excluded from further participation in the study.
- 11. All Subjects must wash out ADHD medications prior to Visit 2. Stimulant ADHD medications (with the exception of study drug), including herbal medications, are prohibited from 5 days prior to Visit 2 for new subjects and prior to Visit 5 for roll-over subjects to the end of the Follow-Up Visit or Early Termination Visit. Before or on the day during the screening period that subjects will need to start the washout of their ADHD medications (for example, 5 days before Visit 2 for stimulants), study site staff will contact the subject's parent/guardian by phone to remind them of the washout ("washout phone call"). Non-Stimulant ADHD medications are prohibited from 14 days prior to the start of the Dose Optimization Phase (Visit 2) to the end of the Follow-Up Visit or Early Termination Visit. Other prohibited medications with their associated time windows when they are prohibited are listed in the protocol.



- 12. KP415 Dose Optimization: Subjects will begin taking open-label KP415 at home the morning following Visit 2. The starting dose of KP415 (Days 1-7 ±3 days) will be 30 mg/day. KP415 dose adjustments, if needed, will be performed at approximately weekly intervals between visits (at Visits 3 and 4). Actual visit dates may deviate from exactly being spaced 7 days apart such that the total duration of the Dose Optimization Phase is 3 weeks (21 days) ±3 days. The daily doses of KP415 used in the Dose Optimization Phase will be 20, 30, and 40 mg (dose optimization range of ≥20 and ≤40 mg). At Visits 3 and 4, based on the CGI scores, interview with the parent/guardian/caregiver, and safety data, the Investigator will evaluate the subject's therapeutic responses and tolerability to treatment and decide whether the current KP415 dose should be increased, decreased, or remain the same for the next week of dosing. If subjects experience symptoms of intolerance during the at-home treatment, they must contact the clinical site, and, at the discretion of the Investigator, their KP415 dose may be adjusted before the next scheduled visit. Unscheduled visits between Visits 2, 3, and 4 are allowed as needed, at the discretion of the Investigator.
- 13. Drug Accountability & Compliance Assessment: All study drug will be recorded by each site's pharmacy staff member or Investigator-delegated employee. A record of the study drug accountability will be prepared and kept by the clinical site.
- 14. ADHD-Rating Scale-5 (ADHD-RS-5) assessment: 1 assessment at the indicated visits.
- 15. Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID): For confirmation of ADHD diagnosis at Screening.
- 16. Clinical Global Impressions—Severity (CGI-S) scale assessment: 1 assessment at the indicated visits.
- 17. Clinical Global Impressions-Improvement (CGI-I) scale assessment: 1 assessment at the indicated visits.
- 18. Children's Sleep Habits Questionnaire (CSHQ) assessment: 1 assessment at Visit 2.
- 19. Adverse Events: To be assessed and recorded in the eCRF following the first dose of open-label drug (KP415), on Day 1, through either Follow-Up or Early Termination. Subject's parent/guardian will be instructed to contact the study site for the reporting of AEs during the dosing periods at home.
- 20. Concomitant Medications: new and/or changed medications and dose, medical treatments and/or therapies will be recorded at Screening through either Follow-Up or Early Termination.
- 21. Actual visit dates in the Dose Optimization Phase may deviate from exactly being spaced 7 days apart such that the total duration of the Dose Optimization Phase ranges between 18 and 24 days (21 ±3 days). Any allowed deviation (up to 3 days in total) of the targeted 21-day Dose Optimization Phase will be carried over into the actual days for the subsequent visits.
- 22. Subjects who meet withdrawal criteria post-dose during the Dose Optimization Phase (after at least one dose of study drug is administered) will complete Early Termination procedures as listed in the Schedule of Events in Table 3. This includes subjects who do not meet the eligibility criteria to continue in the Treatment Phase. At the discretion of the Investigator, ensuring the safety of the subjects, any Early Termination procedures that were already performed on the same day as part of the procedures of the Dose Optimization Phase, do not need to be repeated. Subjects who withdraw early from the study and complete the ET procedures will not return for a Follow-Up Visit. Therefore, the ET Visit is the End-of-Study (EOS) for these subjects.
- 23. The procedures at Screening are different between subjects rolled over from Study KP415.E01 and new subjects. Therefore, the Screening Visit for roll-over subjects is designated as Visit 1B, and for new subjects is designated Visit 1A. Visits 2, 3 and 4 are not needed for subjects rolled over from Study KP415.E01 because their optimum dose was determined in the Dose Optimization Phase of Study KP415.E01. Therefore, roll-over subjects from Study KP415.E01 will start with Visit 1B as the first visit of the current study, followed by Visit 5 as the next visit (roll-over subjects will not have Visits 2, 3 and 4).
- 24. The Screening Visit for roll-over subjects (Visit 1B) may occur on the same day as the EOS (Visit 7, Follow-Up) in Study KP415.E01 or later, and must occur within 30 days before Visit 5 in the current study. For roll-over subjects, the Investigator has the option to use the clinical laboratory (clinical chemistry, hematology and urinalysis) results from the Follow-Up Visit in Study KP415.E01 (Visit 7) in lieu of collecting new blood samples at Screening (Visit 1B) in the current study, as long as the clinical laboratory samples from the E01 study were collected within 30 days prior to Screening (Visit 1B) in the current study. For all roll-over subjects who are children of childbearing potential, a blood sample for the measurement of a serum pregnancy test is needed at Visit 1B. For other assessments required at Visit 1B (C-SSRS, for example), the Visit 7 assessments from the E01 study (if collected) can be used as long as Visit 1B is conducted on the same day as Visit 7 in the E01 study. Visit 7 clinical laboratory samples collected during KP415.E01 (also used as the Visit 1B results) are not required to be collected under fasting conditions. During Visit 1B of the current study, the study site will document whether these samples were collected under fasting/non-fasting conditions, and this will be recorded in the database.



Table 2: Schedule of Events (Treatment Phase [First 6 Months; All Subjects])

| ASSESSMENTS | | | | | | O<br>TREA | OPEN-LABEL TREATMENT PHASE 19 | ABEL PHASE | 19 | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 1-29 | 30 | 31-59 | 09 | 61-89 | 06 | 91- | 120 | 121- | 150 | 151- | 180 |
| Study Day | О | (±5 | (±5 | (±5 | (±5 | (±5 | (±5 | 119 | (±5 | 149 | (±5 | 179 | (±5 |
| for forms | > | Days) | Days) | Days) | Days) | Days) | Days) | (±5<br>Days) | Days) | (±5<br>Days) | Days) | (±5<br>Days) | Days) |
| Visit Number | 5 | | 9 | | 7 | | 8 | | 6 | | 10 | | 11 |
| Inclusion/Exclusion | X | | | | | | | | | | | | |
| Medical History <sup>1</sup> | X | | | | | | | | | | | | |
| Physical Examination <sup>2</sup> | | | | | | | | | | | | | X |
| Body Weight, Height, BMI <sup>3</sup> | X | | X | | X | | X | | X | | X | | X |
| Vital Signs <sup>4</sup> | X | | X | | X | | X | | X | | X | | X |
| 12-Lead ECG <sup>5</sup> | | | | | | | | | | | | | X |
| Chemistry/Hematology/Urinalysis | | | | | | | | | | | | | X |
| Urine MPH Screen (roll-overs) 6 | X | | | | | | | | | | | | |
| Pregnancy Test 7 | X | | X | | X | | X | | X | | X | | X |
| C-SSRS <sup>8</sup> | X | | X | | X | | X | | X | | X | | X |
| Prohibited Medications 9 | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Eligibility Criteria (new subjects) <sup>10</sup> | X | | | | | | | | | | | | |
| Enrollment in Treatment Phase <sup>11</sup> | X | | | | | | | | | | | | |
| Open-Label KP415 Dosing 12 | | X | X | X | X | X | X | X | X | X | X | X | X |
| Drug Accountability & Compliance Assessment | $X^{22}$ | | | | | | | | | | | | × |
| ADHD-RS-5 13 | X | | X | | X | | X | | X | | X | | X |
| CGI-S <sup>14</sup> | X | | X | | X | | X | | X | | X | | X |
| CGI-I 15 | X | | | | | | | | | | | | |
| CSHQ 16 | X | | X | | X | | X | | X | | X | | X |
| Adverse Events <sup>17</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant Medications 18 | X | | X | | × | | × | | X | | X | | X |
| Interim Analysis <sup>23</sup> | | | | | | | | | | | | | X |

EOS = End of Study; ET = Early Termination; BMI = Body Mass Index; ECG = Electrocardiogram; see footnotes for other abbreviations.



Table 3: Schedule of Events (Treatment Phase [Second 6 Months], and Early Termination and Follow-Up Visits [All Subjects])

| ASSESSMENTS | | | | | TRE | OPEN-LABEI<br>ATMENT PHA | OPEN-LABEL TREATMENT PHASE 19 | E 19 | | | | | $\mathbf{ET}^{21}$ (EOS) | $\mathbf{ET}^{21}$ (EOS) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | 181-<br>209<br>(±5<br>days) | 210<br>(±5<br>days) | 211-<br>239<br>(±5<br>days) | 240<br>(±5<br>days) | 241-<br>269<br>(±5<br>days) | 270<br>(±5<br>days) | 271-<br>299<br>(±5<br>days) | 300<br>(±5<br>days) | 301-<br>229<br>(±5<br>days) | 330<br>(±5<br>days) | 331-<br>359<br>(±5<br>days) | 360<br>20<br>(±5<br>days) | 1 | 343-<br>383<br>(±2<br>days) <sup>19</sup> |
| Visit Number | | 12 | | 13 | | 14 | | 15 | | 16 | | 17 | ı | 18 |
| Physical Examination <sup>2</sup> | | | | | | | | | | | | X | X | |
| Body Weight, Height, BMI <sup>3</sup> | | X | | X | | X | | X | | X | | X | X | X |
| Vital Signs <sup>4</sup> | | X | | X | | X | | X | | X | | X | X | X |
| 12-Lead ECG <sup>5</sup> | | | | | | | | | | | | X | X | |
| Chemistry/Hematology/ | | | | | | | | | | | | X | X | |
| conditions) | | | | | | | | | | | | * | * ; | |
| Pregnancy Test 7 | | X | | X | | X | | X | | X | | X | X | X |
| C-SSRS <sup>8</sup> | | X | | X | | X | | X | | X | | X | X | X |
| Prohibited Medications 9 | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Open-Label KP415 Dosing <sup>12</sup> | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Drug Accountability & Compliance Assessment | | X | | X | | X | | X | | X | | X | X | |
| ADHD-RS-5 <sup>13</sup> | | X | | X | | X | | X | | X | | X | | |
| CGI-S <sup>14</sup> | | X | | X | | X | | X | | X | | X | | |
| CGI-I 15 | | | | | | | | | | | | | | |
| CSHQ 16 | | X | | X | | X | | X | | X | | X | | |
| Adverse Events <sup>17</sup> | × | X | X | X | X | X | X | × | X | X | × | × | X | X |
| Concomitant Medications 18 | | X | | X | | X | | X | | X | | X | X | X |

EOS = End of Study; ET = Early Termination; BMI = Body Mass Index; ECG = Electrocardiogram; see footnotes for other abbreviations.

<sup>1.</sup> Medical History: A complete medical history including chronic conditions, relevant surgical procedures (with start date), history of drug and alcohol use. 2. Physical examination at Visit 11, and at Visit 17 (EOT) or at Early Termination (if possible)

<sup>3.</sup> Body weight, height and BMI at each visit. Height will be recorded in centimeters (cm) with the subject's shoes removed. Body weight will be measured in

kilograms (kg); subjects will remain in their normal clothing with shoes and jacket (and/or outer clothing) removed



- diastolic measurements), pulse rate (beats per minute), respiratory rate (breaths per minute), and oral temperature. Vital signs will be collected once at each visit. 4. Vital sign measurements will be obtained after the subject has been seated for at least 3 minutes. Vital signs will include sitting blood pressure (systolic and 5. Electrocardiogram (ECG): A 12-lead ECG will be obtained after the subject has been in the supine position for at least 3 minutes. Abnormal ECGs may be
  - repeated for confirmation in which case only the repeated ECG will be recorded. The QT interval corrected for heart rate will be calculated with Fridericia's
- 6. Urine Screen for Methylphenidate (MPH): Urine samples will be tested for MPH at Visit 5 for roll-over subjects. A urine dipstick (e.g., NarcoCheck®) will be used to screen for the presence of MPH in the urine. All ADHD medications must be washed out by Visit 5 for roll-over subjects. Subjects with a positive MPH urine screen at Visit 5 will be excluded from further participation in the study or may be retested at a later date, and may be enrolled if the MPH urine screen retest is negative as long as the Screening Window is adhered to.
  - 7. A urine pregnancy test will be performed for female subjects of childbearing potential at all visits during the Treatment Phase, and at Early Termination or Follow-Up. A positive pregnancy test before the last dose of study drug will exclude a subject from further participation in the study.
- Termination or Follow-Up. Subjects who have, in the opinion of the Investigator, clinically significant suicidal ideation/behavior, based on history of attempted 8. Columbia Suicide Severity Rating Scale (C-SSRS): The "Children's Since Last Visit" version will be assessed at all visits the Treatment Phase, and at Early 9. Stimulant ADHD medications (with the exception of study drug), including herbal medications, are prohibited from 5 days prior to Visit 5 to the end of the suicide and the C-SSRS assessment at Screening or at any time before the last dose of study drug, will be excluded from further participation in the study Follow-Up Visit or Early Termination Visit.
  - Non-Stimulant ADHD medications are prohibited from 14 days prior to the start of Visit 5 to the end of the Follow-Up Visit or Early Termination Visit. Other prohibited medications with their associated time windows when they are prohibited are listed in the protocol body text.
- Treatment Phase. This is not needed for subjects rolled over from Study KP415.E01 because their optimum dose was determined in the Dose Optimization Phase 10. At Visit 5, for new patients, the Investigator will evaluate the eligibility criteria based on assessments in the Dose Optimization Phase, for continuation into of Study KP415.E01. Rolled-over subjects from Study KP415.E01 will start with Visit 1B as the first visit of the current study, followed by Visit 5 as the next the subsequent Treatment Phase. For subjects eligible for the Treatment Phase, the optimal daily KP415 dose will be used as the daily KP415 dose in the visit (rolled-over subjects will not have Visits 2, 3, and 4).
  - current study. Subjects not rolled over from Study KP415.E01 within 45 days of the last dose of study drug, may be enrolled in the current study as new subjects rolled over from Study KP415.E01 will be enrolled in the Treatment Phase of the current study (Visit 5) within 45 days after the last dose of study drug in Study KP415.E01 (Visit 6 in Study KP415.E01). New subjects will continue to the Treatment Phase immediately after the end of the Dose Optimization Phase in the (they will need to start with Screening and Dose Optimization Phase). At the start of the Treatment Phase (Visit 5), the appropriate open-label study drug to be KP415.E01 (they will need to have completed Study KP415.E01), or at the end of the Dose Optimization Phase in the current study for new subjects. Subjects Treatment Phase. The determination of tolerability and adequate dose-response will be determined in Study KP415.E01 for subjects rolled over from Study 11. Enrollment in the Treatment Phase: Subjects able to tolerate at least 20 mg/day of KP415 and with an adequate dose-response will be enrolled into the taken at home once-a-day in the morning on each of the days of the Treatment Phase until the next visit will be dispensed to the subjects.
    - Based on individual tolerability and dose-response during the Treatment Phase, at the discretion of the Investigator, the KP415 dose may be changed (increased capsule/day) in the morning at home under supervision of their parent or legal guardian. The final dose of study drug will be administered on the last day of the capsule). The dose level is an optimized KP415 dose of 20, 30, or 40 mg determined at the end of the Dose Optimization Phase in Study KP415.E01 for rolledoccur earlier than Day 360 for some or all subjects. Study drug will be taken orally with up to 210-240 mL of water. The capsule needs to be swallowed whole 12. Study Drug Administration: All subjects eligible to participate in the Treatment Phase will receive non-blinded oral capsules with active KP415 drug (one Treatment Phase (Day 360 ±20 days; Visit 17). If the study is stopped earlier based on the stopping rules, the last day of the Treatment Phase (Visit 17) may or decreased, but one of the 3 dose levels of 20, 30, or 40 mg KP415 capsules). All study drugs will be given orally. Subjects will take study drug (one over subjects from Study KP415.E01, or as determined at the end of the Dose Optimization Phase in the current study for new subjects.



(without crushing, cutting, crushing, chewing, opening, or dissolving) or may be taken by sprinkling the contents of the capsule over a small amount of applesauce, or putting the contents in a small amount of water.

- 13. ADHD-Rating Scale-5 (ADHD-RS-5) assessment: 1 assessment at the indicated visits.
- 14. Clinical Global Impressions-Severity (CGI-S) scale assessment: 1 assessment at the indicated visits.
- 15. Clinical Global Impressions-Improvement (CGI-I) scale assessment: 1 assessment at Visit 5 for new subjects only.
  - 16. Children's Sleep Habits Questionnaire (CSHQ) assessment: 1 assessment at the indicated visits.
- 7. Adverse Events: To be assessed and recorded in the eCRF following the first dose of open-label drug (KP415), through either Early Termination or Follow-Up. Subject's parent/guardian will be instructed to contact the study site for the reporting of AEs while away from the study site.
- 18. Concomitant Medications: new and/or changed medications and dose, medical treatments and/or therapies will be recorded at Visit 5 through either Follow-Up or Early Termination.
- 19. To allow flexibility in scheduling visits, actual visit dates for individual subjects in the Treatment Phase may deviate from exactly being spaced 30 days apart (up to 30 ±5 days from the previous visit) such that the total duration of the Treatment Phase may be in the range of 360 ±20 days (340-380 days from Visit 5 to Visit 17). The Follow-Up Visit (3 days after the last dose) therefore falls between Day 343 and Day 383, but has its own window of ±2 days added.
  - 20. The end of the Treatment Phase is on Day 360 ±20 days (Visit 17), after all post-dosing procedures are completed.
- Termination procedures. At the discretion of the Investigator, ensuring the safety of the subjects, any Early Termination procedures that were already performed on the same day as part of the procedures of the Treatment Phase, do not need to be repeated. Subjects who withdraw early from the study and complete the ET 21. Subjects who meet withdrawal criteria post-dose during the Treatment Phase (after at least one dose of study drug is administered) will complete Early procedures will not return for a Follow-Up Visit. Therefore, the ET Visit is the End-of-Study (EOS) for these subjects.
  - delegated employee. A record of the study drug accountability will be prepared and kept by the clinical site at each visit for subjects receiving study drug since the previous visit (including drug accountability at Visit 5 for drug returned from the last week of the Dose Optimization Phase, by new subjects). 22. Drug Accountability & Compliance Assessment: All study drug will be recorded by each site's pharmacy staff member or Investigator-
- and other studies, the Sponsor may stop the study. Treatment in the current study will continue as planned while the interim analysis is conducted. If the decision months) of treatment. After the completion of the interim analysis, based on the acceptance of the clinical and nonclinical safety database from the current study is made to stop the study, all subjects remaining in the study will undergo the EOT Visit (with safety evaluations including fasting safety labs and ECGs) and a 23. An interim analysis of the safety data will be conducted after approximately all subjects remaining in the study have completed 180 days (approximately 6





## 4. Statistical Analysis and Reporting

The analyses contained in this Statistical Analysis Plan will assess the safety and efficacy of KP415 and will be included in the CSR. The final analysis will be performed after database lock when all subjects have been followed through Visit 18 (Days 343-383  $\pm 2$  days), unless the study is stopped early (see Section 4.2 for stopping rules).

The protocol will include an interim analysis after approximately all subjects remaining in the study have completed 180 days (approximately 6 months) of treatment (Visit 11). The focus of the interim analysis will be the safety assessments during the first 6 months of treatment in the Treatment Phase. The table, figure, and listing (TLF) shells that will be used for both the interim and final analyses are contained in this SAP. See Section 4.2 for more details.

#### 4.1. Introduction

Data processing, tabulation of descriptive statistics, calculation of inferential statistics, and graphical representations will be performed primarily using SAS (release 9.4 or higher). If the use of other software is warranted, the final statistical methodology report will detail what software was used for what purposes.

Continuous (quantitative) variable summaries will include the number of subjects (n) with non-missing values, mean, standard deviation (SD), coefficient of variation (CV%), median, minimum, and maximum.

Categorical (qualitative) variable summaries will include the frequency and percentage of subjects who are in the particular category or each possible value, as well as 95% confidence intervals (CIs). In general, the denominator for the percentage calculation will be based upon the total number of subjects in the study population for the treatment, unless otherwise specified. The denominator for by-visit displays will be the number of subjects in the relevant study population and treatment with non-missing data at each visit.

The minimum and maximum will be reported with the same degree of precision (ie, the same number of decimal places) as the observed data. Measures of location (mean and median) will be reported to 1 degree of precision more than the observed data and measures of spread (SD) will be reported to 2 degrees of precision more than the observed data.

Percentages will be presented to 1 decimal place, unless otherwise specified.

Unless otherwise indicated, all statistical tests will be conducted at the 0.05 significance level using 2-tailed tests, and P values will be reported. Corresponding 95% CIs will be presented for statistical tests.

A P value of  $\leq 0.10$  but > 0.05 will be considered evidence of a trend. All formal statistical comparisons for continuous variables will be based on the t-test with unequal variances if data is normally distributed. If data is not normally distributed, the non-parametric Wilcoxon/Mann-Whitney rank-sum test will be used. All formal statistical





comparisons for categorical or binary variables will be based on the Chi-square test or Fisher's exact test. Wilson confidence intervals for binomial proportions and differences in binomial proportions will be computed.

Summaries of disposition and efficacy will be presented overall, by any dose of KP415. For safety summaries presented by treatment, the dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. For the dose optimization phase tables, the optimized dose is presented. If a subject receives a lower dose than planned due to tolerability, this will be mentioned in a footnote.

#### 4.2. Interim Analysis and Data Monitoring

An interim analysis of the safety data will be conducted after approximately all subjects remaining in the study have completed 180 days (approximately 6 months) of treatment (Visit 11). The focus of the interim analysis will be the safety assessments (primary endpoints) during the first 6 months of treatment in the Treatment Phase. The safety data will be analyzed using the same statistical methods as planned for the main analysis after completion of the study. The results from the interim safety analysis will be used to determine whether or not the study can be stopped. All other endpoints (including the secondary endpoints) and assessments will also be analyzed as part of the interim analysis. Tables that will be presented in the interim analysis will be flagged in the table of contents.

The study may be stopped for any of the following reasons, whichever comes first:

- 1. After the completion of the interim analysis, based on the acceptance of the clinical and nonclinical safety database from the current study and other studies, the Sponsor may stop the study. Treatment in the current study will continue as planned while the interim analysis is conducted. If the decision is made to stop the study, all subjects remaining in the study will undergo the EOT Visit (with safety evaluations including fasting safety labs and ECGs) and a Follow-Up Visit.
- 2. After approximately 100 subjects have completed 360 days (approximately 1 year) of treatment. Other subjects remaining in the study (treated at that time for less than 360 days) will undergo the EOT Visit (with safety evaluations including fasting safety labs and ECGs) and a Follow-Up Visit.

#### 5. Analysis Populations

The following analysis populations are planned for this study:

- Treatment-phase Safety Population: The Treatment-phase Safety Population will include all enrolled subjects who received at least 1 dose of study medication in the Treatment Phase and had at least 1 post-dose safety assessment in the Treatment Phase. All baseline and safety data (the latter during the Treatment Phase) will be analyzed using this population.
- **Efficacy Population:** The Efficacy Population will include all enrolled subjects who received at least 30 days of study medication in the Treatment Phase, who had





adequate data to assess the change from baseline of the efficacy parameters, and who had no protocol deviations that could affect the efficacy parameters. All efficacy analyses and sleep behavior results (via CSHQ) across the Treatment Phase will be analyzed using this population.

• Dose-optimization Safety Population: The Dose-optimization Safety Population will include all enrolled subjects in the Dose Optimization Phase ("New Subjects") who received at least one dose of study medication in the Dose Optimization Phase and had at least one post-dose safety assessment in the Dose Optimization Phase. All data from the Dose Optimization Phase will be analyzed using this population.

## 6. General Issues for Statistical Analysis

#### 6.1. Statistical Definitions and Algorithms

#### 6.1.1. Baseline

The baseline for the safety parameters (physical examinations, vital signs, height, weight, BMI, ECG parameters, clinical laboratory tests, and C-SSRS scores) will be the last observation recorded prior to the first dose of study drug. This is measured at either Visit 1A or Visit 2 for new subjects and Visit 1B for roll-over subjects.

The baseline for ADHD-RS-5, CGI-S, and CSHQ will be measured at Visit 5 for roll-over subjects and at Visit 2 for new subjects.

#### **6.1.2.** Adjustments for Covariates

Where statistical modelling is performed, the baseline value of that assessment will be used as a covariate.

#### **6.1.3.** Multiple Comparisons

No adjustments will be made for multiple comparisons; all analyses will be conducted at the  $\alpha = 0.05$  level.

#### 6.1.4. Handling of Dropouts or Missing Data

Subjects who withdraw from the study during the Treatment Phase will not be replaced. Subjects who withdraw from the study during the Dose Optimization Phase may be replaced. Missing data will not be imputed for safety analyses.

For the analysis of efficacy, a sensitivity analysis will be performed in which missing ADHD-RS-5, CGI-S, CGI-I, and CSHQ scores during the Dose Optimization Phase and Treatment Phase will be imputed using Last Observation Carried Forward (LOCF).





## 6.1.5. Analysis Visit Windows

For all analyses, unscheduled and/or repeated measurements will only be included if a scheduled measurement is not available and the unscheduled/repeated measurement falls within the analysis visit windows as described in Table 1, Table 2, and Table 3. Otherwise, visits will be analyzed as scheduled.

#### 6.1.6. Pooling of Sites

Safety and efficacy data will be pooled across all sites. Additionally, subgroup analyses will be performed in which safety, efficacy, and CSHQ endpoints are analyzed by site. See Section 8 and Section 9 for more details.

## 6.1.7. Derived Variables

- ADHD-RS-5 Inattention Subscale Score = summed severity and frequency ratings of the 9 item inattentiveness ADHD rating sub scale. Each item is scored from a range of 0 (reflecting no symptoms or a frequency of never or rarely) to 3 (reflecting severe symptoms or a frequency of very often), so that the subscale score ranges from 0 to 27.
- ADHD-RS-5 Hyperactivity/Impulsivity Subscale Score = summed severity and frequency ratings of the 9 item hyperactivity/impulsivity ADHD rating subscale. Each item is scored from a range of 0 (reflecting no symptoms or a frequency of never or rarely) to 3 (reflecting severe symptoms or a frequency of very often), so that the subscale score ranges from 0 to 27.
- ADHD-RS-5 Total Score = summed severity and frequency ratings of the 18 item ADHD rating scale based on Diagnostic and Statistical Manual of Mental Disorders, 5<sup>th</sup> edition (DSM-5)<sup>4</sup> criteria. Each item/symptom is scored from a range of 0 (reflecting no symptoms or a frequency of never or rarely) to 3 (reflecting severe symptoms or a frequency of very often), so that the total ADHD-RS-5 scores range from 0 to 54.
- Total Sleep Disturbance Score = summed frequency ratings of the 33-item modified, abbreviated CSHQ used to assess examine sleep behavior in small children<sup>5,6</sup>. Items are rated on a 3-point scale of "Usually," "Sometimes," and "Rarely" for occurrences in the following sleep domains: bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep disordered breathing, and daytime sleepiness.
- Change from baseline = value at current time point value at baseline
- Percent change from baseline = (change from baseline / baseline) \* 100. If both baseline and change from baseline are 0 then percent change from baseline will be set to 0.



- TEAE = any adverse event (AE) with an onset date/time between the initiation of study drug and 5 days after the last dose of study drug. This will include any AE with onset prior to initiation of study drug and increased severity after the treatment administration.
- Treatment duration (days) = LASTDAY FIRSTDAY + 1 day

where

LASTDAY is the date of last dose, and

FIRSTDAY is the date of first dose.

- Mean daily dose = sum of all doses taken (in mg) / total number of days from day after previous visit to current visit
- BMI = weight (kg) / [(height (cm)/100) \* (height (cm)/100)]
- Body surface area (BSA) =  $\sqrt{[\text{height(cm)} * \text{weight(kg)}]/3600}$ )
- Treatment compliance = Number of pills taken/Total number of days on the study

Acceptable Compliance is defined as 80-100% (inclusive) of the total pills to be taken on study (eg, 288-360 pills if the subject completes the study).

• Fridericia's correction (QTcF) will be derived as follows:  $QTcF = \frac{QT}{\sqrt[3]{RR}}$ 

where

Relative rate: RR = 60 / HR

HR = Heart rate obtained from the ECG.

#### 6.1.8. Data Adjustments/Handling/Conventions

All collected data will be presented in listings. Data not subject to analysis according to this plan will not appear in any tables or graphs but will be included only in the data listings.

All P values will be displayed in 4 decimals and rounded using standard scientific notation (eg, 0.XXXX). If a P value less than 0.0001 occurs it will be shown in tables as <0.0001.

All AEs and medical histories will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 20.1 thesaurus or higher. Prior and concomitant medications will be coded using the World Health Organization-Drug Dictionary Enhanced (WHO-DDE) version September 2017 or higher.

A treatment related AE is any AE with a relationship to the study drug of possibly, probably, or definitely related.





If partial AE or medication dates occur, the convention for replacing missing dates for the purpose of statistical analysis is as follows:

For partial AE and medication start dates:

- If the year is unknown, then do not impute the date but assign a missing value.
- If the year is known, but the month or month and day is unknown, then:
  - If the year matches the year of first dose date and the end date (if present) is after first dose date, then impute as the month and day of the first dose date.
  - Otherwise, assign 01 January.
- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the first dose date, then impute as the day of the first dose date.
  - o Otherwise, assign 01.

For partial AE and medication end dates:

- If the year is unknown, then do not impute the date but assign as missing value.
- If the year is known, but the month or month and day is unknown, then:
  - o If the year matches the year of the last date of the study (date of last contact if subject lost to follow-up; date of completion or early termination otherwise), then impute as the month and day of the last date of the study.
  - o Otherwise, assign 31 December.
- If the year and month are known, but the day is unknown, then:
  - o If the month and year match the month and year of the last date of the study, then impute as the day of the last date of the study.
  - Otherwise, assign the last day of the month.

#### 7. Study Subjects and Demographics

## 7.1. Disposition of Subjects and Withdrawals

Disposition will include an accounting of the number of subjects enrolled into each treatment, the number of roll-over subjects who participated in KP415.E01, the number of subjects who received treatment, reasons for discontinuation from the study, and number of subjects in each analysis population. For each main reason for early discontinuation, an assessment will be made to determine when in the course of treatment most subjects discontinued early. The last dose received prior to discontinuation will be listed.





The number of subjects remaining in the study by visit will also be presented by treatment.

Percentages will be based on the number of subjects in the Dose-Optimization Safety Population for Visits 2-4 and in the Treatment-Phase Safety Population for Visits 5-18.

Listings of subject disposition and inclusion and exclusion criteria not met will be provided.

#### 7.2. Protocol Violations and Deviations

All protocol deviations will be listed.

## 7.3. Demographics and Other Baseline Characteristics

Summary statistics for age, gender, child-bearing potential, ethnicity, race, height, weight, BSA, and BMI will be presented.

For the continuous variables, the number of non-missing values and the mean, standard deviation, median, minimum and maximum will be tabulated.

For the categorical variables, the counts and percentages of each value will be tabulated.

Baseline variables and dose of study drug will also be presented by study status. Study status will be categorized as "Completed Study" or "Discontinued Early."

The number and percent of subjects reporting various medical histories and prior medications, grouped by MedDRA system organ class and preferred term, will be tabulated.

These analyses will be conducted for the Treatment-Phase Safety Population.

Individual subject listings will be presented for ADHD diagnosis and confirmation as well as the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).

#### 7.4. Exposure and Compliance

At Visit 5, subjects will be dispensed an unblinded bottle with 35 capsules of the optimized dose of KP415 (either 20 mg, 30 mg or 40 mg capsules). For roll-over subjects from Study KP415.E01, the optimized dose as determined in Study KP415.E01 will be used. For new subjects, the optimized dose will be determined at the end of the Dose Optimization Phase in the current study.

Subjects will return to the research clinic at Visits 6-16 with unused study drug, and will be dispensed a new bottle with 35 capsules of either 20 mg, 30 mg, or 40 mg KP415 product. Since the Investigator may increase or decrease the dose of KP415 during the Treatment Phase, based on individual tolerability and dose response, the capsule strengths dispensed at Visit 6 to Visit 16 may be different from the previous visit.

The number of capsules dispensed and returned will be accounted for by site staff. Acceptable compliance is defined as 80-100% (inclusive). The number and percentage of





subjects compliant with study treatment will be tabulated. The total number of doses received as well as the mean, standard deviation, minimum, median and maximum doses received will be tabulated overall and by visit, beginning with Visit 6, the first visit in which study drug is returned.

The mean daily dose of KP415 (mg), the mean daily dose of KP415 by body weight (mg/kg), and the mean daily dose of KP415 by body surface area (mg/m²) will be calculated by visit, and will be compared over time (percent change from starting dose in the Treatment Phase) to show dose changes over the course of the study. The number and percent of subjects who did not take study drug for any continuous period of  $\geq 7, \geq 14$ ,  $\geq 21$ , and  $\geq 28$  days in the Treatment Phase will also be reported.

Results from the capsule swallowing test will be listed.

#### 8. Efficacy Analysis

#### 8.1. Secondary Efficacy Analysis

The secondary efficacy endpoints include changes in ADHD-RS-5, CGI-S, CGI-I, and CSHO.

During the Dose Optimization Phase (new subjects only):

• CGI-S will be assessed at each visit (Screening to Visit 5). ADHD-RS-5 will be administered at Visits 2 through Visit 5. CGI-I will be assessed at Visits 3, 4, and 5 (since CGI-I is an ADHD improvement assessment, it will not be assessed at Screening or at Visit 2).

During the Treatment Phase (all subjects):

• ADHD-RS-5, CSHQ, and CGI-S will be assessed at each visit (Visit 5 to Visit 17, EOT).

Changes in ADHD-RS-5, CGI-S, and CSHQ will be analyzed in the Efficacy Population. Changes in CGI-I will be analyzed in the Efficacy Population during the Dose Optimization Phase. Change in mean scores between baseline and subsequent study visits will be analyzed using a 2-sided paired t-test at a significance level of 0.05. Summary statistics and the 95% confidence interval of the mean will be presented as will the change from baseline and percent change from baseline. Normality assumptions will be tested separately on all evaluable ADHD-RS-5 and CSHQ data across all dose groups using the Shapiro-Wilk and Anderson-Darling methods. If both P values for the normality tests are >0.01, the data for that particular outcome will be considered normally distributed. Otherwise, if one or both P values are  $\leq$ 0.01, the data for that particular outcome will be considered non-normal and then the null hypothesis that the median change from baseline is 0 will be tested with the Wilcoxon signed rank test.

Change from baseline and percent change from baseline will be summarized by overall subjects. The analyses will be repeated in the Dose-Optimization Safety population for new subjects. No statistical inference will be performed for this analysis population.

Categorical CGI-S and CGI-I results will be summarized by study visit.





Section 6.1.7 describes the derivations of the above variables and their baseline values.

Subgroup analyses will be performed for the Treatment Phase by gender, age, duration of treatment, race, study site, previous stimulant exposure and treatment. Mean and SD change from baseline ADHD-RS-5 /CSHQ score for each subgroup will be displayed for each visit. Duration of treatment and age will be broken up into quartiles. If the distribution of duration of treatment or age is such that the use of quartiles does not lead to distinct intervals of values, other cut points will be examined (e.g. tertiles, above/below median). CGI-S results will also be presented for the above subgroups.

#### 9. Safety and Tolerability Analysis

Safety will be evaluated from reported AEs, physical exam results, and changes in the following: clinical laboratory values, vital signs, height, weight, BMI, ECG, and C-SSRS scores.

Descriptive statistics will be calculated for quantitative safety data and frequency counts and percentages will be compiled for classification of qualitative safety data. Individual subject listings will be prepared for all safety data.

The primary safety analyses will be performed on the Treatment-Phase Safety Population. Data from the Dose-Optimization Safety Population will be summarized descriptively. All safety data will be presented in the listings.

#### 9.1. Adverse Events

Adverse events with new onset during the study between the initiation of study drug and 5 days after the last dose of study drug will be considered as TEAEs. This will include any AE with onset prior to initiation of study drug and increased severity after the treatment initiation. For AEs occurring on the date of the first dose of study drug, if the time of onset is missing, the AE will be assumed to be treatment emergent.

All AEs, TEAEs, and SAEs will be coded using MedDRA version 20.1 or higher.

The causal relationship of the AE to the study drug is determined by the investigator as Unrelated, Possibly Related, Probably Related, and Definitely Related. These can be mapped to Unrelated (*Unrelated*) and Related (*Possibly Related*, *Probably Related*, and *Definitely Related*).

Adverse event severity grades are reported on a 5-point scale of Grade 1 (*Mild*), Grade 2 (*Moderate*), Grade 3 (*Severe*), Grade 4 (*Life-threatening consequences*), or Grade 5 (*Death related to AE*).

The number and percentage of subjects who experience a TEAE along with the 95% Wilson confidence interval (CI) will be presented.

Summaries of incidence rates (frequencies and percentages) of individual TEAEs will be summarized by MedDRA system organ class (SOC) and preferred term (PT) for overall





subjects and by average dose. This will include overall incidence rates (regardless of severity and relationship to study drug). Such summaries will also be displayed for TEAEs by maximum severity and relationship to study drug. If a particular event is missing the severity and/or relationship, then the severity or relationship will be presented as missing.

Each subject will be counted only once within each SOC and PT. If a subject experiences more than 1 TEAE within a particular SOC and PT, the TEAE with the strongest relationship or the maximum severity, as appropriate, will be included in the summaries of relationship and severity.

Incidences will be presented by descending frequency of SOC and PT within SOC, and then alphabetically within PT where the incidence is the same; this is based on overall subjects.

Missing and partially missing AE start and/or stop dates will be imputed, for the purpose of statistical analysis, according to the specifications described in Section 6.1.8.

In the AE data listings, all AEs will be displayed. Any AEs that are treatment emergent will be flagged.

Subgroup analyses of safety will be performed by gender, age, duration of treatment, race, study site, previous stimulant exposure, and treatment. Duration of treatment and age will be broken up into quartiles. If the distribution of duration of treatment or age is such that the use of quartiles does not lead to distinct intervals of values, other cut points will be examined (e.g. tertiles, above/below median). Subgroup analyses will be performed on the Treatment-Phase Safety Population.

#### 9.1.1. Adverse Events Leading to Withdrawal

A summary of incidence rates (frequencies and percentages) of TEAEs leading to discontinuation of study drug, by average dose, SOC, and PT will be prepared for the Treatment-Phase Safety Population. No inferential statistical tests will be performed.

A data listing of AEs leading to withdrawal of study drug will also be provided, displaying details of the event(s) captured on the CRF.

#### 9.1.2. Deaths and Serious Adverse Events

Any deaths that occured during the study will be listed.

Serious adverse events will be listed and also tabulated by SOC and PT and presented by treatment.

## 9.1.3. Other Significant Adverse Events

In accordance with the 2017 FDA Guidance for Industry<sup>7</sup>, Assessment of Abuse Potential of Drugs<sup>8</sup>, abuse-related AEs will be analyzed in the Treatment Phase using the following MedDRA Preferred Terms:





- Euphoria-related terms: Euphoric mood; Elevated mood; Feeling abnormal; Feeling drunk; Feeling of relaxation; Dizziness; Thinking abnormal; Hallucination; Inappropriate affect
- Terms of altered attention, cognition and mood: Somnolence; Mood disorders and disturbances
- Dissociative/psychotic terms: psychosis; aggression; confusion and disorientation
- Related terms not captured elsewhere: drug tolerance; habituation; drug withdrawal syndrome; substance-related disorders.

The number and percentage of subjects with at least 1 abuse-related AE will be presented. Abuse-related AEs will be categorized by SOC and PT and tabulated by treatment, age, and gender. Age will be broken up into quartiles. If the distribution of age is such that the use of quartiles does not lead to distinct intervals of values, other cut points will be examined (e.g. tertiles, above/below median).

Abuse-related AEs will be flagged in the individual subject listings to show the incident that led to the AEs, the time at which AEs appear following drug administration, the duration of the AEs, and which AEs overlap temporally.

## 9.2. Clinical Laboratory Evaluations

Safety clinical hematology laboratory evaluations will include measures of red blood cell count, white blood cell count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), hemoglobin, hematocrit and platelets, Prothrombin Time (PT) and Partial Thromboplastin Time (PTT).

Serum chemistry laboratory evaluations will include measures of aspartate aminotransferase (AST), alanine aminotransferase (ALT), albumin, alkaline phosphatase, bicarbonate, total bilirubin, blood urea nitrogen, phosphorus (inorganic) calcium, chloride, creatinine phosphokinase, creatinine, gamma glutamyl transferase, glucose, lactate dehydrogenase, potassium, sodium, total protein, thyroid stimulating hormone (TSH), and uric acid. TSH will be measured at Screening only, for new subjects only who did not previously participate in Study KP415.E01.

Urinalysis will include microanalysis for specific gravity, pH, protein, glucose, ketones, blood, nitrites, and leukocytes.

Safety laboratory tests will be summarized as observed values and by post-treatment change from baseline for each of the parameters using descriptive statistics overall at each visit. Categorical urinalysis results will be summarized using frequencies by visit. Shifts from baseline for clinical laboratory values below, within, or above the normal range will be provided for hematology, chemistry, and urinalysis results by visit and treatment. See Section 6.1.1 for the definition of baseline.

Subjects with significant laboratory abnormalities will be identified in data listings. If any laboratory tests are collected at an unscheduled visit post-baseline, the results will be included in listings.

Pregnancy test results and urine screens for alcohol and drugs of abuse will be listed.





## 9.3. Vital Signs

Descriptive summaries of observed values and change from baseline will be calculated for systolic blood pressure, diastolic blood pressure, pulse rate, respiratory rate, and oral temperature by visit and average dose.

Weight, height, BMI, and BSA will be summarized by observed values and by post-treatment change from baseline by visit and treatment.

#### 9.4. Electrocardiograms

A 12-lead ECG will be obtained after the subject has been in a supine position for a minimum of 3 minutes. Abnormal ECGs may be repeated for confirmation in which case only the repeated ECG will be recorded. The QT interval corrected for heart rate will be calculated with Fridericia's formula (QTcF). ECGs will be obtained at Screening, after approximately 6 months of treatment (Visit 11), after the last dose of study drug (Visit 17, EOT), and at Early Termination (if possible). ECG recordings will be evaluated by skilled readers operating from a centralized ECG laboratory.

The number and percentage of subjects with normal, abnormal clinically significant, and abnormal not clinical significant ECG results will be summarized for the Treatment-Phase Safety Population by visit.

## 9.5. Further Safety Evaluations

Suicidal ideation will be assessed by the C-SSRS, Pediatric Version<sup>9</sup>. The "Children's Baseline/Screening" version will be assessed at Screening, and the "Children's Since Last Visit" version will be assessed at all visits of the Dose Optimization Phase (new subjects only), at all of the Treatment Phase visits, and at Follow-Up or Early Termination. For the continuous suicidal ideation, intensity of ideation, and suicidal behavior variables, the number of non-missing values and the mean, standard deviation, minimum, median and maximum will be tabulated by dose and visit. For the categorical variables, the counts and percentages of each value will be tabulated by dose and visit.

A complete physical examination will be completed at Screening, after approximately 6 months of treatment (Visit 11), after the last dose of study drug (Visit 17, EOT), and at Early Termination (if possible). The following body systems will be assessed: general appearance, skin, head, neck, eyes, ears, nose, mouth, and throat (HEENT), lymph nodes, thyroid, musculoskeletal/extremities, cardiovascular system, lungs, abdomen and a brief examination of the neurological system. Physical examination findings will be presented in individual subject listings.

#### 9.6. Concomitant Medication

Summaries of medications that were started prior to dosing and continuing at the time of dosing as well as medications that were starting during dosing or during follow up will be presented using counts and percentages by WHO Drug Anatomical Therapeutic Chemical





(ATC) codes level 4 and level 5 (PT) and treatment for subjects in the Treatment-Phase Safety population.

Individual subject listings will be presented for all concomitant medications, lifetime history of ADHD treatment, and ADHD medication washout.

## 10. Changes from Planned Analysis

Not Applicable

## 11. Other Planned Analysis

Not Applicable





#### 12. References

- 1. US Federal Register. (1998) International Conference on Harmonization; Guidance on Statistical Principles for Clinical Trials. Department of Health and Human Services: Food and Drug Administration [Docket No. 97D-0174]. Federal Register Volume 63, Number 179, pages 49583-49598. September 16, 1998.
- 2. ASA. (2016) Ethical Guidelines for Statistical Practice. Prepared by the Committee on Professional Ethics, April 2016. http://www.amstat.org/about/ethicalguidelines.cfm
- 3. RSS. (2014) The Royal Statistical Society: Code of Conduct, 2014. http://www.rss.org.uk/Images/PDF/join-us/RSS-Code-of-Conduct-2014.pdf.
- 4. American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). Arlington, VA, American Psychiatric Association, 2013.
- 5. Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep, 2000a; 23(8):1043–51.
- 6. Owens J, Spirito A, McGuinn M, Nobile C. Sleep habits and sleep disturbance in schoolaged children. Journal of Developmental and Behavioral Pediatrics, 2000b; 21(1):27-36.
- 7. Food and Drug Administration, Assessment of Abuse Potential of Drugs. (2017, January). Guidance for Industry, U.S. Department of Health and Human Services, Center for Drug Evaluation and Research, Washington, DC.
- 8. Sellers EM, Romach MK. Categorization of Abuse Potential-Related Adverse Events. Clin Pharmacol Drug Dev. 2017 Oct 11. doi: 10.1002/cpdd.394. [Epub ahead of print].
- 9. Posner K, Brent D, Lucas C, Gould M, Stanley B, Brown G, Fisher P, Zelazny J, Burke A, Oquendo M, Mann J. Columbia-Suicide Severity Rating Scale (C-SSRS) Pediatric Baseline Version. New York, NY: The Research Foundation for Mental Hygiene, Inc., 2010.

#### 13. Tables, Listings, and Figures

All listings, tables, and graphs will have a header showing the sponsor company name and protocol and a footer showing the version of SAS, the file name and path, and the source of the data (CRF page or listing number).

#### 13.1. Planned Table Descriptions

The following are planned summary tables for protocol number KP415.S01. The table numbers and page numbers are place holders only and will be determined when the tables are produced.



**Table 4: Demographic Data Summary Tables and Figures** 

| Number | Population | Title |
|---|---|---|
| Table 14.1.1 | All Subjects | Summary of Subject Disposition by Treatment |
| Table 14.1.2 | All Subjects | Summary of Subject Attrition by Treatment |
| Table 14.1.3.1 | Treatment-<br>Phase Safety | Summary of Demographics and Baseline Characteristics by Treatment |
| Table 14.1.3.2 | Treatment-<br>Phase Safety | Summary of Demographics and Baseline Characteristics by<br>Treatment and Study Status |
| Table 14.1.4 | Treatment-<br>Phase Safety | Incidence of Medical Histories by SOC, PT, and Treatment |
| Table 14.1.5.1 | Treatment-<br>Phase Safety | Summary of Prior Medications by ATC Class Level 4, PT, and Treatment |
| Table 14.1.6.1 | Treatment-<br>Phase Safety | Summary of Study Drug Compliance by Treatment and Visit |
| Table 14.1.6.2 | Treatment-<br>Phase Safety | Summary of Mean Daily Doses by Visit |
| Table 14.1.6.3 | Treatment-<br>Phase Safety | Summary of Missed Doses by Treatment |

# 13.2. Efficacy Data

**Table 5: Efficacy Data** 

| Number | Population | Title |
|---|---|---|
| Table 14.2.1.1.1 | Efficacy | Summary of ADHD-RS-5 Scores by Study Visit |
| Table 14.2.1.1.2 | Efficacy | Summary of ADHD-RS-5 Scores by Study Visit Using Imputation |
| Table 14.2.1.1.3 | Efficacy | Summary of ADHD-RS-5 Scores by Study Visit and Gender |
| Table 14.2.1.1.4 | Efficacy | Summary of ADHD-RS-5 Scores by Study Visit and Age |
| Table 14.2.1.1.5 | Efficacy | Summary of ADHD-RS-5 Scores by Study Visit and Duration of Treatment |
| Table 14.2.1.1.6 | Efficacy | Summary of ADHD-RS-5 Scores by Study Visit and Race |
| Table 14.2.1.1.7 | Efficacy | Summary of ADHD-RS-5 Scores by Study Visit and Site |
| Table 14.2.1.1.8 | Efficacy | Summary of ADHD-RS-5 Scores by Study Visit and Previous Stimulant Exposure |
| Table 14.2.1.1.9 | Efficacy | Summary of ADHD-RS-5 Scores by Study Visit and Treatment |
| Table 14.2.1.2.1 | Efficacy | Summary of CGI-S by Study Visit |
| Table 14.2.1.2.2 | Efficacy | Summary of CGI-S by Study Visit and Gender |
| Table 14.2.1.2.3 | Efficacy | Summary of CGI-S by Study Visit and Age |



| Number | Population | Title |
|---|---|---|
| Table 14.2.1.2.4 | Efficacy | Summary of CGI-S by Study Visit and Duration of Treatment |
| Table 14.2.1.2.5 | Efficacy | Summary of CGI-S by Study Visit and Race |
| Table 14.2.1.2.6 | Efficacy | Summary of CGI-S by Study Visit and Site |
| Table 14.2.1.2.7 | Efficacy | Summary of CGI-S by Study Visit and Previous Stimulant Exposure |
| Table 14.2.1.2.8 | Efficacy | Summary of CGI-S by Study Visit and Treatment |
| Table 14.2.1.3.1 | Efficacy | Summary of CGI-I by Study Visit |
| Table 14.2.1.4.1 | Efficacy | Summary of CSHQ Total Sleep Disturbance Score by Study Visit |
| Table 14.2.1.4.2 | Efficacy | Summary of CSHQ Total Sleep Disturbance Score by Study Visit Using Imputation |
| Table 14.2.1.4.3 | Efficacy | Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Gender |
| Table 14.2.1.4.4 | Efficacy | Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Age |
| Table 14.2.1.4.5 | Efficacy | Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Duration of Treatment |
| Table 14.2.1.4.6 | Efficacy | Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Race |
| Table 14.2.1.4.7 | Efficacy | Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Site |
| Table 14.2.1.4.8 | Efficacy | Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Previous Stimulant Exposure |
| Table 14.2.1.4.9 | Efficacy | Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Treatment |



# 13.3. Safety Data

# **Table 6: Safety Data**

| Number | Population | Title |
|---|---|---|
| 14.3.1 Displays of A | Adverse Events | |
| Table 14.3.1.1.1 | Treatment-Phase<br>Safety | Summary of Treatment Emergent Adverse Events by Treatment |
| Table 14.3.1.1.2 | Dose-<br>Optimization<br>Safety | Summary of Treatment Emergent Adverse Events by Treatment |
| Table 14.3.1.2.1 | Treatment-Phase<br>Safety | Incidence of Treatment Emergent Adverse Events by SOC, PT, and Treatment |
| Table 14.3.1.2.2 | Dose-<br>Optimization<br>Safety | Incidence of Treatment Emergent Adverse Events by SOC, PT, and Treatment |
| Table 14.3.1.3.1 | Treatment-Phase<br>Safety | Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Treatment |
| Table 14.3.1.3.2 | Dose-<br>Optimization<br>Safety | Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Treatment |
| Table 14.3.1.3.3 | Treatment-Phase<br>Safety | Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Gender |
| Table 14.3.1.3.4 | Treatment-Phase<br>Safety | Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Age |
| Table 14.3.1.3.5 | Treatment-Phase<br>Safety | Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Duration of Treatment |
| Table 14.3.1.3.6 | Treatment-Phase<br>Safety | Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Race |
| Table 14.3.1.3.7 | Treatment-Phase<br>Safety | Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Site |
| Table 14.3.1.3.8 | Treatment-Phase<br>Safety | Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Previous Stimulant Exposure |
| Table 14.3.1.4.1 | Treatment-Phase<br>Safety | Incidence of Treatment Related Treatment Emergent Adverse Events by SOC, PT, and Treatment |
| Table 14.3.1.4.2 | Dose-<br>Opimization<br>Safety | Incidence of Treatment Related Treatment Emergent Adverse Events by SOC, PT, and Treatment |
| Table 14.3.1.5.1 | Treatment-Phase<br>Safety | Incidence of Treatment Emergent Adverse Events Leading to Study<br>Drug Discontinuation by SOC, PT, and Treatment |



| Number | Population | Title |
|---|---|---|
| Table 14.3.1.5.2 | Dose-<br>Optimization<br>Safety | Incidence of Treatment Emergent Adverse Events Leading to Study<br>Drug Discontinuation by SOC, PT, and Treatment |
| 14.3.2 Summary of Deaths, Other Serious and Significant Adverse Events | | |
| Table 14.3.2.1 | Treatment-Phase<br>Safety | Incidence of Serious Adverse Events by SOC, PT, and Treatment, |
| Table 14.3.2.2 | Dose-<br>Optimization<br>Safety | Incidence of Serious Adverse Events by SOC, PT, and Treatment |
| 14.3.3 Narratives of I | Deaths, Other Seri | ous and Certain Other Significant Adverse Events |
| Table 14.3.3.1.1 | Treatment-Phase<br>Safety | Listing of Adverse Events Leading to Study Drug Discontinuation |
| Table 14.3.3.1.2 | Dose-<br>Optimization<br>Safety | Listing of Adverse Events Leading to Study Drug Discontinuation |
| Table 14.3.3.2.1 | Treatment-Phase<br>Safety | Listing of Serious Adverse Events |
| Table 14.3.3.2.2 | Dose-<br>Optimization<br>Safety | Listing of Serious Adverse Events |
| Table 14.3.3.3.1 | Treatment-Phase<br>Safety | Listing of Deaths |
| Table 14.3.3.3.2 | Dose-<br>Optimization<br>Safety | Listing of Deaths |
| Table 14.3.3.4.1 | Treatment-Phase<br>Safety | Incidence of Abuse Related Adverse Events by SOC, PT, and Treatment |
| Table 14.3.3.4.2 | Treatment-Phase<br>Safety | Incidence of Abuse Related Adverse Events by SOC, PT, and Age |
| Table 14.3.3.4.3 | Treatment-Phase<br>Safety | Incidence of Abuse Related Adverse Events by SOC, PT, and Gender |
| Table 14.3.3.4.4 | Dose-<br>Optimization<br>Safety | Incidence of Abuse Related Adverse Events by SOC, PT, and Treatment |
| 14.3.4 Abnormal Laboratory Value | | |
| NA | | |
| 14.3.5 Laboratory Data Summary Tables | | |
| Table 14.3.5.1.1 | Treatment-Phase<br>Safety | Summary of Hematology Laboratory Results by Study Visit and Treatment |



| Number | Population | Title |
|---|---|---|
| Table 14.3.5.1.2 | Treatment-Phase<br>Safety | Shift from Baseline in Hematology Laboratory Results by Study Visit and Treatment |
| Table 14.3.5.2.1 | Treatment-Phase<br>Safety | Summary of Serum Chemistry Laboratory Results by Study Visit and Treatment |
| Table 14.3.5.2.2 | Treatment-Phase<br>Safety | Shift from Baseline in Serum Chemistry Laboratory Results by Study<br>Visit and Treatment |
| Table 14.3.5.3.1 | Treatment-Phase<br>Safety | Shift from Baseline in Quantitative Urinalysis Laboratory Results by Study Visit and Treatment |
| Table 14.3.5.3.2 | Treatment-Phase<br>Safety | Shift from Baseline in Quantitative Urinalysis Laboratory Results by<br>Study Visit and Treatment |
| Table 14.3.5.3.3 | Treatment-Phase<br>Safety | Summary of Qualitative Urinalysis Laboratory Results by Study Visit and Treatment |
| 14.3.6 Other Safety Data Summary Tables | | |
| Table 14.3.6.1 | Treatment-Phase<br>Safety | Summary of Vital Signs by Study Visit, and Treatment |
| Table 14.3.6.2.1 | Treatment-Phase<br>Safety | Summary of 12-Lead Electrocardiogram by Study Visit and Treatment |
| Table 14.3.6.2.2 | Treatment-Phase<br>Safety | Summary of 12-Lead Electrocardiogram Interpretation by Study Visit and Treatment |
| Table 14.3.6.3 | Treatment-Phase<br>Safety | Summary of Columbia-Suicide Severity Rating Scale (C-SSRS) |
| Table 14.3.6.4 | Treatment-Phase<br>Safety | Summary of Concomitant Medications by ATC Class Level 4, PT, and Treatment |





## 13.4. Other Data Summary Tables

## 13.5. Planned Listing Descriptions

The following are planned data and patient/subject data listings for protocol number KP415.S01.

In general, one listing will be produced per CRF domain. All listings will be sorted by treatment, site, and subject number. All calculated variables will be included in the listings.

In all listings a blank line will be placed between each subject. Within a data listing, if an item appears line after line (eg, repetition of subject number), then only the first occurrence will be displayed.

In data listings, the information for one subject will be kept on one page if at all possible, rather than splitting a subject's information across pages.

**Table 7: Planned Listings** 

| Number | Population | Title / Summary |
|---|---|---|
| 16.2.1 Subject Dis | continuations/Com | pletions |
| Listing 16.2.1 | All Subjects | Subject Disposition |
| 16.2.2 Protocol De | eviations | |
| Listing 16.2.2.1 | All Subjects | Inclusion and Exclusion Criteria Not Met |
| Listing 16.2.2.2 | All Subjects | Protocol Deviations |
| 16.2.3 Subjects Ex | cluded from the E | fficacy Analyses |
| Listing 16.2.3 | All Subjects | Analysis Populations |
| 16.2.4 Demograph | ic Data and Other | Baseline Characteristics |
| Listing 16.2.4.1 | All Subjects | Demographics and Baseline Information |
| Listing 16.2.4.2 | All Subjects | Medical History |
| Listing 16.2.4.3 | All Subjects | ADHD Diagnosis and Confirmation |
| Listing 16.2.4.4 | All Subjects | Mini International Neuropsychiatric Interview for Children and<br>Adolescents (MINI-KID) |
| 16.2.5 Compliance | e and/or Drug Cone | centration Data |
| Listing 16.2.5.1 | All Subjects | Capsule Swallowing Test |
| Listing 16.2.5.2 | All Subjects | Study Drug Dispensation and Return |
| 16.2.6 Individual Efficacy Response Data | | |
| Listing 16.2.6.1 | All Subjects | ADHD-Rating Scale-5 |
| Listing 16.2.6.2 | All Subjects | Clinical Global Impression (CGI) – Severity |
| Listing 16.2.6.3 | All Subjects | Clinical Global Impression (CGI) – Improvement |


| Number | Population | Title / Summary |
|---|---|---|
| Listing 16.2.6.4 | All Subjects | Children's Sleep Habits Questionnaire |
| 16.2.7 Adverse Even | t Listings (by Subject | et) |
| Listing 16.2.7.1 | All Subjects | Adverse Events |
| 16.2.8 Laboratory V | alues and Other Cli | nical Observations and Measurements (by Subject) |
| Listing 16.2.8.1.1 | All Subjects | Clinical Laboratory Data: Hematology |
| Listing 16.2.8.1.2 | All Subjects | Clinical Laboratory Data: Serum Chemistry |
| Listing 16.2.8.1.3 | All Subjects | Clinical Laboratory Data: Urinalysis |
| Listing 16.2.8.1.4 | All Subjects | Clinical Laboratory Data: Urine Drug Screen and Pregnancy Tests |
| Listing 16.2.8.2 | All Subjects | Vitals Signs |
| Listing 16.2.8.3 | All Subjects | 12-Lead Electrocardiogram (ECG) |
| Listing 16.2.8.4 | All Subjects | Columbia-Suicide Severity Rating Scale (C-SSRS) |
| Listing 16.2.8.5 | All Subjects | Physical Examination |
| Listing 16.2.8.6 | All Subjects | Prior and Concomitant Medications |
| Listing 16.2.8.7 | All Subjects | Lifetime History of ADHD Treatment |
| Listing 16.2.8.8 | All Subjects | ADHD Medication Washout |



**premier** research



Not Applicable



# Tables, Listings, and Listing Shells

# Standard Layout for all Tables, Listings, and Figures 13.7.

The following standard layout will be applied to all Tables, Listings, and Figures in support of this study. Note that programming notes may be added if appropriate after each TLF shell.



# Figure 1: Standardized Layout

| KemPharm, Inc. | Page xx of xx |
|---|---|
| Protocol: KP415.S01 | Version |
| <table, figure="" listing,=""> xx.x.x</table,> | |
| <title figure="" listing="" of="" or="" table="">&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Study Population and if applicable subgroup Description&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Body of Table, Listing or Figure&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;&lt;Note: If directly Applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote 1 &lt;if applicable&gt; Recommendation is to keep footnotes to a minimum&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote 2 &lt;i&gt;&lt;if applicable&gt;&lt;/i&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote n &lt;if applicable&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;tr&gt;&lt;td&gt;Footnote n+1 &lt;pre&gt;pgm path and name&gt;, &lt;date&gt;&lt;/pre&gt;&lt;/td&gt;&lt;td&gt;&lt;/td&gt;&lt;/tr&gt;&lt;/tbody&gt;&lt;/table&gt;</title> | |





#### Planned Table Shells 13.8.

premier



| | KP415 |
|--------------------------------------------------------------|-------------|
| Status | (N=XX) |
| Enrolled | × |
| Study Populations: | |
| Treatment-Phase Safety Population [1] | XX (XX.X%) |
| Efficacy Population [2] | XX (XX.X%) |
| Dose-Optimization Safety Population [3] | XX (XX.X%) |
| Completed Study | (%X:XX) XX |
| Ongoing in Study | XX (XX.X%) |
| Prematurely Discontinued from Study | XX (XX.X%) |
| Subject withdrawal of consent | XX (XX.X%) |
| Non-compliance with study procedures | XX (XX.X%) |
| Adverse event | XX (XX.X%) |
| Lack of efficacy | XX (XX.X%) |
| Protocol deviation | XX (XX.X%) |
| Lost to follow-up | XX (XX.X%) |
| Sponsor request for early termination of study | XX (XX.X%) |
| Positive pregnancy test | XX (XX.X%) |
| Out-of-range vital signs | XX (XX.X%) |
| Sponsor planned study stop | XX (XX.X%) |
| Other | XX (XX.X%) |
| Participated in KP415.E01 and enrolled as roll-over subjects | XX (XX.X%) |
| | XX (XX. X%) |

Note: Percentages are n/Number of subjects in enrolled \*100. Subjects are summarized overall.
[1] The Treatment-Phase Safety Population includes all subjects who are enrolled in the Treatment Phase and received at least 1 dose of study medication

in the Treatment Phase and had at least 1 post-dose safety assessment in the Treatment Phase.

<sup>[2]</sup> The Efficacy Population includes all enrolled subjects who received at least 30 days of study medication in the Treatment Phase and had adequate data

to assess the change from baseline of the efficacy parameters and no protocol deviations that could affect the efficacy parameters.

[3] The Dose-Optimization Population includes all subjects who are enrolled in the Dose Optimization Phase and received at least 1 dose of study medication in the Dose Optimization Phase and had at least 1 post-dose safety assessment in the Dose Optimization Phase.

SOURCE: Listings 16.2.1, 16.2.3



Table 14.1.2 Summary of Subject Attrition by Study Phase All Subjects

| KP415<br>(N=XX) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) | (%x x x x x x x x x x x x x x x x x x x | XX (XX.X%) |
|---|---|---|---|---|
| Visit Number | Screening Phase:<br>Visit 01A (New Subjects)<br>Visit 01B (Rollover Subjects) | Dose Optimization Phase:<br>Visit 02 (New Subjects)<br>Visit 03 (New Subjects)<br>Visit 04 (New Subjects) | Treatment Phase: | Follow up:<br>Visit 18 |

Note: Percentages are n/Number of subjects in enrolled\*100. Subjects are summarized overall. SOURCE: Listings 16.2.1



Table 14.1.3.1 Summary of Demographics and Baseline Characteristics Treatment-Phase Safety Population

| KP415<br>(N=XX) | XX XX (XX.XX) XX.XX XX.XX XX.XX XX.XX | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | (%X X%)<br>XX (XX X%) |
|---|---|---|---|---|---|
| Variable<br>Statistic or Category | Age (years) n Mean (SD) CV% Median Min, Max | Gender<br>Male<br>Female | Child-Bearing Potential? [1]<br>Yes<br>No | Ethnicity<br>Hispanic or Latino<br>Not Hispanic or Latino | Race<br>American-Indian or Alaska Native<br>Asian<br>Black or African-American<br>Native Hawaiian or Other Pacific Islander<br>White<br>Other<br>More than One Race |

Abbreviations: CV% = coefficient of variation; SD = standard deviation.

Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Subjects are summarized overall.

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Treatment-Phase Safety Population. SOURCE: Listing 16.2.4.1



Table 14.1.3.1 (cont.)
Demographics and Baseline Characteristics
Treatment-Phase Safety Population

| KP415<br>(N=XX) | XX (XX.XX) XX.XX XX.XX XX.X XX.X | XX.X(XX.XX) XX.XX XX.XX XX.XX XX.X | XX.X(XX.XX) XX.XX XX.XX XX.XX XX.XX XX.XX | xx xx<br>xx.xx<br>xx.xx<br>xx.x<br>xx, xx |
|---|---|---|---|---|
| Variable<br>Statistic or Category | Height (cm) n Mean (SD) CV% Median Min, Max | Weight (kg) n Mean (SD) CV% Median Min, Max | Body Surface Area (mg/m²)<br>n<br>Mean (SD)<br>CV%<br>Median<br>Min, Max | Body Mass Index (kg/m²)<br>n<br>Mean (SD)<br>CV%<br>Median<br>Min, Max |

Abbreivations: CV% = coefficient of variation; SD = standard deviation.

Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Subjects are summarized overall.

[1] Only captured for female subjects; percentages are based on the number of female subjects in the Treatment-Phase Safety Population. SOURCE: Listing 16.2.4.1





Table 14.1.3.2
Demographics and Baseline Characteristics by Study Status
Treatment-Phase Safety Population

#### (Same Shell as Table 14.1.3.1)

Programming Note: Update Note to read "Percentages are n/Number of subjects in the Treatment-Phase Safety Population for each study status\*100." Add Listing 16.2.3 to SOURCE. Add a header row that says "Study Status: XXXX", where XXXX is "Completed Study" or "Discontinued Early".

Sponsor KemPharm, Inc. Protocol Number KP415.S01 PCN Number KEMP7419 Statistical Analysis Plan,

**premier** research

Incidence of Medical Histories by SOC and PT Treatment-Phase Safety Population Table 14.1.4

| System Organ Class | KP415 |
|---------------------------------------------------|-------------|
| Preferred Term | (N=XX) |
| Subjects with at least 1 Recorded Medical History | XX (XX.X%) |
| System Organ Class 1 | XX (XX.X%) |
| Preferred Term 1 | XX (XX.X%) |
| Preferred Term 2 | XX (XX.X%) |
| Preferred Term 3 | XX (XX.X%) |
| System Organ Class 2 | XX (XX. X%) |
| Preferred Term 1 | XX (XX. X%) |
| Preferred Term 2 | XX (XX. X%) |
| Preferred Term 3 | XX (XX. X%) |

Abbreviations: PT = Preferred Term; SOC = System Organ Class.

Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Subjects are summarized overall. Medical histories were coded using MedDRA version 20.1. Subjects were counted once for each system organ class (SOC) and once for each preferred term (PT). Medical history terms are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT.

SOURCE: Listing 16.2.4.2

Programming note: SOC & PT text should be in proper case in table, as shown in the shell.

Statistical Analysis Plan, Sponsor KemPharm, Inc. Protocol Number KP415.S01 PCN Number KEMP7419

**premier** research



| ATC Class Level 4<br>Preferred Term (ATC Class Level 5) | KP415<br>(N=XX) |
|---|---|
| Subjects with at least 1 Prior Medication | XX (XX.X%) |
| ATC Class 1 Preferred Term 1 Preferred Term 2 Preferred Term 3 | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |
| ATC Class 2 Preferred Term 1 Preferred Term 2 Preferred Term 3 | XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%)<br>XX (XX.X%) |

using WHO-DDE version September 2017. Prior medications are all medications that were started before the date of the first dose of study drug in the Treatment Phase. Medications are displayed by descending frequency of Anatomic Therapeutic Chemical (ATC) Level 4 classification, by Preferred Term (PT) within ATC, and then alphabetically. Subjects were counted only once for each ATC and PT. SOURCE: Listing 16.2.9.6 Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Subjects are summarized overall. Medications were coded Abbreviations: ATC = Anatomic Therapeutic Chemical; PT = Preferred Term

Programming note: ATC & PT text should be in proper case in table, as shown in the shell.



Summary of Study Drug Compliance by Visit Treatment-Phase Safety Population Table 14.1.6.1

| KP415<br>(N=XX) | XX (XX.X%)<br>XX (XX.X%) | XX XX (XX.XX) XX.XX XX.XX XX.XX XX.XX | XX XX (XX.XX) XX.XX XX.XX XX.X XX.X | XX.X(XX.XX) XX.XX XX.XX XX.XX XX.XX |
|---|---|---|---|---|
| Statistic / Category | Compliant [1]<br>Not Compliant | Total Number of Doses Taken<br>n<br>Mean (SD)<br>CV%<br>Median<br>Min, Max | Total Number of Doses Taken Visit 6<br>n<br>Mean (SD)<br>CV%<br>Median<br>Min, Max | Total Number of Doses Taken Visit 7<br>n Mean (SD)<br>CV%<br>Median<br>Min, Max |

#### Continue for Visits 8-17

Abbreviations: CV% = coefficient of variation; SD = Standard Deviation.

Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Subjects are summarized overall. Number of doses taken is calculated as the number of expected doses (number of days on study, where number of days on study is derived as last treatment – first treatment + 1) minus total number of missed doses, as collected in the CRF.

[1] Subjects were to receive one dose in the morning each day. Acceptable compliance is defined as 80-100% (inclusive) and is derived as number of doses faken / number of expected doses \* 100%. SOURCE: Listing 16.2.5.2



Table 14.1.6.2 Summary of Mean Daily Doses by Visit Treatment-Phase Safety Population

| Study Visit | | Mean Daily Dose (mg)<br>(N = XX) | ng) | Mean Daily I | Mean Daily Dose by Body Weight (mg/kg)<br>(N = XX) | eight (mg/kg) | Mean Da | Mean Daily Dose by BSA ( $mg/m^2$ )<br>(N = XX) | . (mg/m²) |
|---|---|---|---|---|---|---|---|---|---|
| Statistic | Observed | CFB | %CFB | Observed | CFB | %CFB | Observed | CFB | %CFB |
| Visit 5 | | | | | | | | | |
| _ | × | ı | ı | × | ŀ | ŀ | × | 1 | 1 |
| Mean (SD) | XX.X (X.XX) | | | XX.X (X.XX) | | | XX.X (X.XX) | | |
| CV% | XX:XX | | | XX:XX | | | XX:XX | | |
| Median | X.X | | | X:X | | | ×:× | | |
| Min, Max | ×× | | | ×<br>×<br>× | | | XX, XX | | |
| Visit 6 | | | | | | | | | |
| _ | × | × | × | × | × | × | × | × | × |
| Mean | XX.X (X.XX) | XX.X (X.XX) | XX.X (X.XX) | XX.X (X.XX) | XX.X (X.XX) | XX.X (X.XX) | XX.X (X.XX) | XX.X (X.XX) | XX.X (X.XX) |
| %\S | XX:XX | XX:XX | XX:XX | XX:XX | XXX | XXX | XXX | XXX | ××× |
| Median | XX | XXX | XX.X | XXX | ××× | ××× | XXX | ××× | XX.X |
| Min, Max | ××× | ×,× | XX, XX | ××× | ××× | ×, × | ×,× | ××× | ××× |
| | | | 2 | the the the second | oticity Mainie | | | | |
| | | | COUNT | continue for the the remaining visits. | allilly visits. | | | | |

Abbreviations: BSA = body surface area; CFB = change from baseline; CV% = coefficient of variation; SD = standard deviation. Note: Mean daily dose = sum of all doses taken (in mg) / total number of days from the day after the previous visit to current visit. SOURCE: Listing 16.2.5.2



Summary of Missed Doses by Treatment Treatment-Phase Safety Population Table 14.1.6.3

| KP415 | (XX=N) | XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) |
|---|---|---|
| | Number of Days Study Drug Not Taken [1] | ≥7 Days<br>≥14 Days<br>≥21 Days<br>≥28 Days |

Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Subjects are summarized overall. A subject contributes to row if they did not take study drug for the continuous period of specified days.
[1] Subjects were to receive one dose in the morning each day.
SOURCE: Listing 16.2.5.2



Summary of ADHD-RS-5 Scores by Study Visit **Efficacy Population** Table 14.2.1.1.1

Parameter: ADHD-RS-5 Total Score

| | | KP415 | |
|------------------|--------------|--------------|--------------|
| Study Visit | | (N=XX) | |
| Statistic | Observed | CFB | %CFB |
| Baseline [1] | | | |
| | × | × | × |
| Mean (SD) | (XX:XX) | XX:X (XX:XX) | XX.X (XX.XX) |
| (95% ČI of Mean) | (XXX, XXX) | (XX:X, XX:X) | (XXX, XXXX) |
| ČV% | XXXX | XXXX | XXXX |
| Median | ××× | XXX | ××× |
| Min, Max | ×××× | XX, XX | ××× |
| Visit 2 | | | |
| <b>L</b> | × | × | × |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| (95% ČI of Mean) | (XXX, XXX) | (XXX XXXX) | (XXX, XXXX) |
| ČV% | XX.XX | XX.XX | XX:XX |
| Median | XXX | ××× | XXX |
| Min, Max | ××× | ××× | ××× |
| P-value [2] | | XXXXX | |

Abbreviations: CFB = change from baseline; CV% = coefficient of variation; SD = standard deviation.

Note: ADHD-RS-5 Inattention Subscale Score = summed severity and frequency ratings of the 9 item inattentiveness ADHD rating sub scale.

ADHD-RS-5 Hyperactivity/Impulsivity Subscale Score = summed severity and frequency ratings of the 9 item hyperactivity/impulsivity ADHD symptoms or a frequency of very often), so that the subscale scores range from 0 to 27, ADHD-RS-5 Total Score = summed severity and frequency ratings of the 18 item ADHD rating scale (Inattention and Hyperactivity/Impulsivity subscales combined). The total ADHD-RS-5 scores range from 0 to 54. A negative change indicates improvement. 95% Wilson Cls are presented. rating subscale. Each item is scored from a range of 0 (reflecting no symptoms or a frequency of never or rarely) to 3 (reflecting severe

[1] The baseline is measured before the first dose of study drug at Visit 2 for new subjects and at Visit 5 for roll-over subjects. Visit 3 and Visit 4 will only be populated for new subjects in the Dose Optimization Phase. Visits 5-17 will include all subjects in the Treatment Phase.

[2] P-value for testing mean change from baseline to subsequent visit is 0 is calculated using a paired t-test. SOURCE: Listing 16.2.6.1



Summary of ADHD-RS-5 Scores by Study Visit Table 14.2.1.1.1 (cont.) **Efficacy Population** 

Parameter: ADHD-RS-5 Total Score

| | | KP415 | |
|------------------|--------------|--------------|--------------|
| Study Visit | | (XX=N) | |
| Statistic | Observed | CFB | %CFB |
| Visit 4 | | | |
| _ | × | × | × |
| Mean (SD) | XX:X (XX:XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| (95% ČI of Mean) | (XX.X, XX.X) | (XX.X, XX.X) | (XX.X, XX.X) |
| ČV% | XX.XX | XXXX | XX.XX |
| Median | XXX | XXX | ××× |
| Min, Max | ××× | XX, XX | ×,× |
| P-value | | XXXXX | |

Continue for Study Visits 5-17. Repeat for the following parameters: ADHD-RS-5 Inattention Subscale Score; ADHD-RS-5 Housing Visits 5-17. Repeativity/Impulsivity Subscale Score.

Note: ADHD-RS-5 Inattention Subscale Score = summed severity and frequency ratings of the 9 item inattentiveness ADHD rating sub scale. Abbreviations: CFB = change from baseline; CV% = coefficient of variation; SD = standard deviation.

ADHD-RS-5 Hyperactivity/Impulsivity Subscale Score = summed severity and frequency ratings of the 9 item hyperactivity/impulsivity ADHD symptoms or a frequency of very often), so that the subscale scores range from 0 to 27. ADHD-RS-5 Total Score = summed severity and frequency ratings of the 18 item ADHD rating scale (Inattention and Hyperactivity/Impulsivity subscales combined). The total ADHD-RS-5 scores range from 0 to 54. A negative change indicates improvement. 95% Wilson Cls are presented. rating subscale. Each item is scored from a range of 0 (reflecting no symptoms or a frequency of never or rarely) to 3 (reflecting severe

[1] The baseline is measured before the first dose of study drug at Visit 2 for new subjects and at Visit 5 for roll-over subjects. Visit 3 and Visit 4 will only be populated for new subjects in the Dose Optimization Phase. Visits 5-17 will include all subjects in the Treatment Phase.

[2] P-value for testing mean change from baseline to subsequent visit is 0 is calculated using a paired t-test. SOURCE: Listing 16.2.6.1

Programming note: Check assumptions for normality per Section 8.1 of the SAP. If normality assumptions are violated, use the Wilcoxon signed rank test and update the footnote accordingly



Summary of ADHD-RS-5 Scores by Study Visit Using Imputation Efficacy Population (Same shell as Table 14.2.1.1.) Table 14.2.1.1.2

**Programming note**: Add the following footnote "Missing scores were inputed using Last Observation Carried Forward (LOCF)"

Table 14.2.1.1.3 Summary of ADHD-RS-5 Scores by Study Visit and Gender Efficacy Population

(Same shell as Table 14.2.1.1.1)

Programming note: Each subgroup will have its own set of columns. Add 16.2.4.1 to SOURCE.

Table 14.2.1.1.4 Summary of ADHD-RS-5 Scores by Study Visit and Age **Efficacy Population** 

(Same shell as Table 14.2.1.1.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Check cut points per Section 8.1 of SAP. Add 16.2.4.1 to SOURCE. Table 14.2.1.1.5 Summary of ADHD-RS-5 Scores by Study Visit and Duration of Treatment Efficacy Population

(Same shell as Table 14.2.1.1.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Check cut points per Section 8.1 of SAP. Add 16.2.5.2 to SOURCE. 



Table 14.2.1.1.6 Summary of ADHD-RS-5 Scores by Study Visit and Race Efficacy Population

# (Same shell as Table 14.2.1.1.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Add 16.2.4.1 to SOURCE.

Table 14.2.1.1.7 Summary of ADHD-RS-5 Scores by Study Visit and Site Efficacy Population

# (Same shell as Table 14.2.1.1.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Add 16.2.1 to SOURCE.

Table 14.2.1.1.8 Summary of ADHD-RS-5 Scores by Study Visit and Previous Stimulant Exposure Efficacy Population

### (Same shell as Table 14.2.1.1.1)

Programming note: Each subgroup will have its own set of columns (subgroups include Previous Stimulant Exposure and No Stimulant Exposure). Add 16.2.8.6 to SOURCE. Table 14.2.1.1.9 Summary of ADHD-RS-5 Scores by Study Visit and Treatment Efficacy Population

# (Same shell as Table 14.2.1.1.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Add footnote "Treatment groups are based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented." Add 16.2.5.2 to SOURCE.



Table 14.2.1.2.1 Summary of CGI-S by Study Visit Efficacy Population

| Study Visit | 3 N | KP415<br>(N=XX) |
|-------------------------------------------|-------------|-----------------|
| Statistic | (%) u | 95% CI |
| Screening [1] | × | |
| 0 = Not Assessed | XX (XX.X%) | (XX.X%, XX.X%) |
| 1 = Normal, Not at All III | XX (XX.X%) | (XX.X%, XX.X%) |
| 2 = Borderline Mentally III | XX (XX:X%) | (XX.X%, XX.X%) |
| 3 = Mildly III | XX (XX:X%) | (XX.X%, XX.X%) |
| 4 = Moderately III | XX (XX.X%) | (XX.X%, XX.X%) |
| 5 = Markedly III | XX (XX.X%) | (XX.X%, XX.X%) |
| 6 = Severely III | XX (XX.X%) | (XX.X%, XX.X%) |
| 7 = Among the Most Extremely III Patients | (XX.X%) | (XX.X%, XX.X%) |
| Baseline [2] | × | |
| 0 = Not Assessed | XX (XX.X%) | (XX.X%, XX.X%) |
| 1 = Normal, Not at All III | (%X:X%) | (XX.X%, XX.X%) |
| 2 = Borderline Mentally III | XX (XX.X%) | (XX.X%, XX.X%) |
| 3 = Mildly III | XX (XX:X%) | (XX.X%, XX.X%) |
| 4 = Moderately III | (%X:X%) | (XX.X%, XX.X%) |
| 5 = Markedly III | XX (XX: X%) | (XX.X%, XX.X%) |
| 6 = Severely III | (%X:X%) | (XX.X%, XX.X%) |
| 7 = Among the Most Extremely III Patients | XX (XX.X%) | (XX.X%, XX.X%) |

#### Repeat for Visits 3-17

Abbreviation: CGI-S = Clinical Global Impression – Severity; CI = confidence interval.

Note: Percentages are n/Number of subjects in the Efficacy Population at each visit\*100. The CGI-S rates the severity of the subject's illness at the time of assessment, relative to the clinician's past experience with subjects who have the same diagnosis. Subjects are summarized by treatment recieved. 95% Wilson CIs are presented.

[1] Screening will only include new subjects at Visit 01A. [2] The baseline is measured before the first dose of study drug at Visit 2 for new subjects and at Visit 5 for roll-over subjects. Visit 3 and Visit 4 will only be populated for new subjects in the Dose Optimization Phase. Visits 5-17 will include all subjects in the Treatment Phase.

SOURCE: Listing 16.2.6.2



Table 14.2.1.1.2 Summary of CGI-S by Study Visit by Study Visit and Gender Efficacy Population

# (Same shell as Table 14.2.1.2.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Change SOURCE to Listing 16.2.6.2. Add 16.2.4.1 to SOURCE.

Table 14.2.1.2.3 Summary of CGI-S by Study Visit and Age Efficacy Population

# (Same shell as Table 14.2.1.2.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Check cut points per Section 8.1 of SAP. Change SOURCE to Listing 16.2.6.2. Add 16.2.4.1 to SOURCE.

Table 14.2.1.2.4 Summary of CGI-S by Study Visit and Duration of Treatment Efficacy Population

#### (Same shell as Table 14.2.1.2.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Check cut points per Section 8.1 of SAP. Change SOURCE to Listing 16.2.6.2. Add 16.2.5.2 to SOURCE. Table 14.2.1.2.5

Table 14.2.1.2.5 Summary of CGI-S by Study Visit and Race Efficacy Population

# (Same shell as Table 14.2.1.2.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup.

Change SOURCE to Listing 16.2.6.2. Add 16.2.4.1 to SOURCE.



Table 14.2.1.2.6 Summary of CGI-S by Study Visit and Site Efficacy Population

# (Same shell as Table 14.2.1.2.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Change SOURCE to Listing 16.2.6.2. Add 16.2.1 to SOURCE.

Table 14.2.1.2.7 Summary of CGI-S by Study Visit and Previous Stimulant Exposure Efficacy Population

# (Same shell as Table 14.2.1.2.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Change SOURCE to Listing 16.2.6.2. Add 16.2.8.6 to SOURCE.

Table 14.2.1.2.8 Summary of CGI-S by Study Visit and Treatment Efficacy Population

### (Same shell as Table 14.2.1.2.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Change SOURCE to Listing 16.2.6.2. Add 16.2.5.2 to SOURCE.



Summary of CGI-I by Study Visit Efficacy Population Dose Optimization Phase (New Subjects Only) Table 14.2.1.3.1

| | $\overline{A}$ | P415 |
|------------------------|----------------|----------------|
| Study Visit | Z) | (X=XX) |
| Statistic | l (%) | 95% CI |
| Visit 3 | × | |
| 0 = Not Assessed | XX (XX.X%) | (XX:X%, XX:X%) |
| 1 = Very Much Improved | XX (XX.X%) | (XX:X%, XX:X%) |
| 2 = Much Improved | XX (XX.X%) | (XX.X%, XX.X%) |
| 3 = Minimally Improved | XX (XX.X%) | (XX:X%, XX:X%) |
| 4 = No Change | XX (XX.X%) | (XX.X%, XX.X%) |
| 5 = Minimally Worse | XX (XX.X%) | (XX:X%, XX:X%) |
| 6 = Much Worse | XX (XX.X%) | (XX.X%, XX.X%) |
| 7 = Very Much Worse | XX (XX.X%) | (XX.X%, XX.X%) |

#### Continue for Visit 4 and Visit 5

Abbreviation: CGI-I = Clinical Global Impression – Improvement; CI = confidence interval.

Note: Percentages are n/Number of subjects in the Efficacy Population at each visit\*100. The CGI-I measures the overall improvement in the subject's condition post-treatment. The Investigator will rate the subject's total improvement whether or not it is due entirely to drug treatment. By definition, all CGI-I assessments are evaluated against baseline conditions. Subjects are summarized by treatment received. 95% Wilson CIs are presented.

SOURCE: Listing 16.2.6.3



Table 14.2.1.4.1 Summary of CSHQ Total Sleep Disturbance Score by Study Visit Efficacy Population

# (Same shell as Table 14.2.1.1.1)

Programming note: Add CSHQ = Children's Sleep Habits Questionnaire to abbreviations in footnote. Change SOURCE to Listing 16.2.6.4.

Table 14.2.1.4.2
Summary of CSHQ Total Sleep Disturbance Score by Study Visit Using Imputation Efficacy Population

# (Same shell as Table 14.2.1.1.1)

Programming note: Add CSHQ = Children's Sleep Habits Questionnaire to abbreviations in footnote. Add the following footnote "Missing scores were inputed using Last Observation Carried Forward (LOCF)". Change SOURCE to Listing 16.2.6.4.

Table 14.2.1.4.3 Summary of CSHQ Total Sleep Disturbance Score by Study Visit by Study Visit and Gender Efficacy Population

#### (Same shell as Table 14.2.1.1.1)

Programming note: Add CSHQ = Children's Sleep Habits Questionnaire to abbreviations in footnote. Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Change SOURCE to Listing 16.2.6.4. Add 16.2.4.1 to SOURCE. Table 14.2.1.4.4 Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Age

# Efficacy Population

(Same shell as Table 14.2.1.1.1)

Programming note: Add CSHQ = Children's Sleep Habits Questionnaire to abbreviations in footnote. Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Check cut points per Section 8.1 of SAP. Change SOURCE to Listing 16.2.6.4. Add 16.2.4.1 to SOURCE




Table 14.2.1.4.5
Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Duration of Treatment
Efficacy Population

#### (Same shell as Table 14.2.1.1.1)

Programming note: Add CSHQ = Children's Sleep Habits Questionnaire to abbreviations in footnote. Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Check cut points per Section 8.1 of SAP. Change SOURCE to Listing 16.2.6.4. Add 16.2.5.2 to SOURCE.

Table 14.2.1.4.6 Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Race Efficacy Population

## (Same shell as Table 14.2.1.1.1)

Programming note: Add CSHQ = Children's Sleep Habits Questionnaire to abbreviations in footnote. Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Change SOURCE to Listing 16.2.6.4. Add 16.2.4.1 to SOURCE. Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Site Table 14.2.1.4.7

# Efficacy Population

(Same shell as Table 14.2.1.1.1)

Programming note: Add CSHQ = Children's Sleep Habits Questionnaire to abbreviations in footnote. Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Change SOURCE to Listing 16.2.6.4. Add 16.2.1 to SOURCE.

Table 14.2.1.4.8
Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Previous Stimulant Exposure Efficacy Population

#### (Same shell as Table 14.2.1.1.1)

Programming note: Add CSHQ = Children's Sleep Habits Questionnaire to abbreviations in footnote. Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Change SOURCE to Listing 16.2.6.4. Add 16.2.8.6 to SOURCE.



Table 14.2.1.4.9 Summary of CSHQ Total Sleep Disturbance Score by Study Visit and Treatment Efficacy Population

# (Same shell as Table 14.2.1.1.1)

Programming note: Add CSHQ = Children's Sleep Habits Questionnaire to abbreviations in footnote. Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Change SOURCE to Listing 16.2.6.4. Add 16.2.5.2 to SOURCE.



Summary of Treatment Emergent Adverse Events by Treatment Treatment-Phase Safety Population Table 14.3.1.1.1

| | | KP415 | | | |
|---|---|---|---|---|---|
| | 20 mg<br>(N=XX) | 30 mg<br>(N=XX) | 40 mg<br>(N=XX) | ÓΞ | Overall<br>(N=XX) |
| Category | (%) u | (%) u | (%) u | (%) u | 95% CI |
| Subjects with at least 1 TEAE | XX (XX.X%) | (%X:X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Maximum Severity of TEAE<br>Grade 1 | (XX:XX) | (%X:X%) | (%X:XX) | (XX.X%) | (XX:X%; XX:X%) |
| Grade 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Grade 3 | XX (XX.X%) | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Grade 4 | XX (XX.X%) | (%X:XX) XX | (%X:XX) XX | XX (XX.X%) | (XX.X%, XX.X%) |
| Grade 5 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Subjects with a Related TEAE [2] | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Subjects with a TEAE Leading to Discontinuation of Study Drug | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Subjects with an SAE | (%X:XX) XX | (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Subjects with an AE leading to Death | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |

MedDRA version 20.1. A TEAE is any AE with an onset date/time between the initiation of study drug and 5 days after the last dose of study drug. This will include any AE with onset prior to initiation of study drug and increased severity after the treatment administration. 95% Wilson CIs are presented.
[1] Related TEAEs are those marked as Possibly Related, Probably Related, or Definitely Related on the CRF.
SOURCE: Listing 16.2.7.1 Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Treatment groups are based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. AEs were coded using Abbreviations: CI = confidence interval; CRF = Case Report Form; TEAE = Treatment emergent adverse event; SAE = Serious adverse event.

Programming note: Ensure correct MedDRA version is printed in footnote. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add "16.2.5.2" to the SOURCE line.





Summary of Treatment Emergent Adverse Events by Treatment Dose-Optimization Safety Population Table 14.3.1.1.2

Programming Note: Update footnote with Dose-Optimization Safety Population. Since treatment groups presented are based on the optimized dose (mg) from the Dose Optimization Phase, actual doses need to be determined from the data. Update footnote to read "Treatment groups are based on treatment received. The optimized dose is presented."



Incidence of Treatment Emergent Adverse Events by SOC, PT, and Treatment Treatment-Phase Safety Population Table 14.3.1.2.1

| System Organ Class (N=XX) | | | | | |
|---|---|---|---|---|---|
| | 20 mg | 30 mg | 40 mg | ŏ | Overall |
| | (N=XX) | (N=XX) | (XX=N) | <b>Z</b> ) | (X=XX) |
| | (%) u | (%) u | n (%) | (%) u | 95% CI |
| Subjects with at least 1 TEAE XX (XX.X%) | ( (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| System Organ Class 1 XX (XX.X%) | ( (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| | (XX.XX) | XX (XX.X%) | (%X:XX) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Preferred Term 2 XX (XX. X%) | (XX.XX) | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (XX:X%, XX:X%) |
| Preferred Term 3 XX (XX.X%) | (XX.X%) | (%X:X%) XX | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| System Organ Class 1 XX (XX.X%) | ( (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Preferred Term 1 XX (XX. X% | (%X:XX) | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Preferred Term 2 XX (XX.X%) | (XX.XX) | XX (XX.X%) | (%X:X%) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Preferred Term 3 XX (XX. X% | (XX.X%) | XX (XX.X%) | XX (XX.X%) | (%X:X%) XX | (XX.X%, XX.X%) |

version 20.1. A TEAE is any AE with an onset date/time between the initiation of study drug and 5 days after the last dose of study drug. This will include any AE with onset prior to initiation of study drug and increased severity after the treatment administration. Subjects are counted once for each SOC and once for each PT. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. 95% Wilson CIs are presented.

SOURCE: Listing 16.2.7.1 beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. AEs were coded using MedDRA Abbreviations: CI = confidence interval; PT = Preferred Term; SOC = System Organ Class; TEAE = treatment emergent adverse event.

Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Treatment groups are based on treatment received. The dose received at the

Programming note: SOC & PT text should be in proper case in table, as shown in the shell. Ensure correct MedDRA version is printed in footnote. Since treatment groups presented are based on the dose (mg) received at the beginning of the treatment-phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add "16.2.5.2" to the SOURCE line.



Table 14.3.1.2.2 Incidence of Treatment Emergent Adverse Events by SOC, PT, and Treatment Dose-Optimization Safety Population

## (Same Shell as Table 14.3.1.2.1)

Programming note: Update footnote with Dose-Optimization Safety Population. Since treatment groups presented are based on the optimized dose (mg) from the Dose Optimization Phase, actual doses need to be determined from the data. Update footnote to read "Treatment groups are based on treatment received. The optimized dose is presented."



Table 14.3.1.3.1 Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Treatment Treatment-Phase Safety Population

| | | KP415 | | | |
|---|---|---|---|---|---|
| System Organ Class<br>Preferred Term | 20 mg<br>(N=XX) | 30 mg<br>(N=XX) | 40 mg<br>(N=XX) | δŻ | Overall (N=XX) |
| Maximum Severity | (%) u | (%) u | (%) u | n (%) | 95% CI |
| Subjects with at least 1 TEAE | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Any Event (Total) | | | | | |
| Mild | (%X:XX)<br>XX | (%X:XX)<br>XX | (%X:XX)<br>XX | (%X:XX)<br>XX | (XX.X%, XX.X%) |
| Moderate | (%X XX)<br>XX (XX XX) | XX (XX.X%)<br>XX (XX.X%) | (%X XX) XX | (XX XX)<br>XX (XX X%) | (XX.X%, XX.X%)<br>(XX.X%, XX.X%) |
| Life-threatening consequences | (%X:XX)<br>XX | (%X;XX)<br>XX (XX;XX) | (%X:XX)<br>(%X:XX)<br>(%X:XX) | (%X:XX)<br>XX (XX:X%) | (%X:XX:%X:XX) |
| Death related to AE | (%X:X%)<br>XX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| System Organ Class 1<br>Any Event (Total) | | | | | |
| Mild | XX (XX.X%) | (%X:XX) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Moderate | (%X:X%)<br>XX | (%X:XX) XX | (%X:X%)<br>XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Severe | (%X:X%)<br>XX | (%X:XX) XX | (%X:X%)<br>XX | (%X:XX) | (XX.X%, XX.X%) |
| Life-threatening consequences | XX (XX.X%) | (%X:XX) XX | (%X:X%)<br>XX | (%X:X%) | (XX.X%, XX.X%) |
| Death related to AE | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Missing | XX (XX X%) | XX (XX.X%) | XX (XX.X%) | (%X.XX) | (XX.X%, XX.X%) |
| Preferred Term 1<br>Mild | XX (XX: X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| : | | | | | |

version 20.1. A TEAE is any AE with an onset date/time between the initiation of study drug and 5 days after the last dose of study drug. This will include any AE with onset prior to initiation of study drug and increased severity after the treatment administration. Subjects are counted once for each SOC and once for each PT. The severity shown is the greatest severity reported for a particular subject (Death related to AE > Life-threatening consequences > Severe > Moderate > Mild). AEs with a missing severity were counted as Missing. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. 95% Wilson CIs are presented. Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Treatment groups are based on treatment received. The dose received at the beginning of the Treatment Phase, is presented. AEs were coded using MedDRA Abbreviations: CI = confidence interval; PT = Preferred Tem; SOC = System Organ Class; TEAE = treatment emergent adverse event.

Programming note: SOC & PT text should be in proper case in table, as shown in the shell. Ensure correct MedDRA version is printed in footnote. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add "16.2.5.2" to the SOURCE line.

SOURCE: Listing 16.2.7.1



Table 14.3.1.3.2 Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Treatment Dose-Optimization Safety Population

# (Same shell as Table 14.3.1.3.1)

Programming note: Update footnote with Dose-Optimization Phase Safety Population. Since treatment groups presented are based on the optimized dose (mg) from the Dose-Optimization Phase, actual doses need to be determined from the data. Update footnote to read "Treatment groups are based on treatment received. The optimized dose is presented."

Table 14.3.1.3.3 Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Gender Treatment-Phase Safety Population

#### (Same shell as Table 14.3.1.3.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Add 16.2.4.1 to SOURCE.

Table 14.3.1.3.4 Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Age Treatment-Phase Safety Population

#### (Same shell as Table 14.3.1.3.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Add 16.2.4.1 to SOURCE.

Table 14.3.1.3.5 Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Duration of Treatment Treatment-Phase Safety Population

#### (Same shell as Table 14.3.1.3.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Add 16.2.5.2 to SOURCE.



Table 14.3.1.3.6 Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Race Treatment-Phase Safety Population

#### (Same shell as Table 14.3.1.3.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Add 16.2.4.1 to SOURCE.

Table 14.3.1.3.7 Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Site Treatment-Phase Safety Population

#### (Same shell as Table 14.3.1.3.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Add 16.2.1 to SOURCE.

Table 14.3.1.3.8 Incidence of Treatment Emergent Adverse Events by Maximum Severity, SOC, PT, and Previous Stimulant Exposure Treatment-Phase Safety Population

#### (Same shell as Table 14.3.1.3.1)

Programming note: Each subgroup will have its own set of columns. If there are too many subgroups such that the table would be too wide, repeat the table for each subgroup. Add 16.2.8.6 to SOURCE.



Table 14.3.1.4.1 Incidence of Treatment Related Adverse Events by SOC, PT, and Treatment Treatment-Phase Safety Population

| | | KP415 | | | |
|---|---|---|---|---|---|
| | 20 mg | 30 mg | 40 mg | ð | Overall |
| System Organ Class | (X=X) | (XX=N) | (X=X) | Ξ) | (N=XX) |
| Preferred Term | (%) u | n (%) | n (%) | (%) u | 95% CI |
| Subjects with at least 1 Treatment Related<br>TEAE | (%X:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Preferred Term 1 | XX (XX: X%) | (%X:X%) XX | XX (XX.X%) | (%X:X%) XX | (XX.X%, XX.X%) |
| Preferred Term 2 | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Preferred Term 1 | | (%X:X%) XX | (%X:XX) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Preferred Term 2 | (%X:X%) | (%X:XX) XX | (%X:XX) XX | (%X:X%) | (XX.X%, XX.X%) |
| Preferred Term 3 | (%X:X%) | (%X:X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |

Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Treatment groups are based on treatment received. The dose received at the Abbreviations: CI = confidence interval; PT = Preferred Tem; SOC = System Organ Class; TEAE = treatment emergent adverse event.

beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. AEs were coded using MedDRA version 20.1. A TEAE is any AE with an onset date/time between the initiation of study drug and 5 days after the last dose of study drug. This will include any AE with onset prior to initiation of study drug and increased severity after the treatment administration. A treatment related TEAE is an AE that is marked as being possibly, probably, or definitely related to treatment. Subjects are counted once for each SOC and once for each PT. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by

PT. 95% Wilson Cls are presented. SOURCE: Listing 16.2.7.1

Programming note: SOC & PT text should be in proper case in table, as shown in the shell. Ensure correct MedDRA version is printed in footnote. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add "16.2.5.2" to the SOURCE line.





Incidence of Treatment Related Adverse Events by SOC, PT, and Treatment Dose-Optimization Safety Population (Same Shell as Table 14.3.1.4.1) Table 14.3.1.4.2

Programming note: Update footnote with Dose-Optimization Safety Population. Since treatment groups presented are based on the optimized dose (mg) from the Dose Optimization Phase, actual doses need to be determined from the data. Update footnote to read "Treatment groups are based on treatment received. The optimized dose is presented."



Table 14.3.1.5.1 Incidence of Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by SOC, PT, and Treatment Treatment-Phase Safety Population

#### (Same shell as Table 14.3.1.2.1)

Incidence of Treatment Emergent Adverse Events Leading to Study Drug Discontinuation by SOC, PT, and Treatment Dose-Optimization Safety Population Table 14.3.1.5.2

## (Same shell as Table 14.3.1.2.1)

Programming note: Update footnote with Dose-Optimization Safety Population. Since treatment groups presented are based on the optimized dose (mg) from the Dose Optimization Phase, actual doses need to be determined from the data. Update footnote to read "Treatment groups are based on treatment received. The optimized dose is presented."

Table 14.3.2.1 Incidence of Serious Adverse Events by SOC, PT, and Treatment Treatment-Phase Safety Population

### (Same shell as Table 14.3.1.2.1)

Table 14.3.2.2 Incidence of Serious Adverse Events by SOC, PT, and Treatment Dose-Optimization Safety Population

#### (Same shell as Table 14.3.1.2.1)

Programming note: Update footnote with Dose-Optimization Safety Population. Since treatment groups presented are based on the optimized dose (mg) from the Dose Optimization Phase, actual doses need to be determined from the data. Update footnote to read "Treatment groups are based on treatment received. The optimized dose is presented."


Table 14.3.3.1.1
Listing of Adverse Events Leading to Study Drug Discontinuation
Treatment-Phase Safety Population

| Subject<br>ID | Treatment [1] | System Organ Class/<br>Preferred Term/<br>Verbatim Term | Start Date/Time (Study Day)/ Severity/<br>End Date/Time (Study Day) Relationship | Severity/<br>Relationship | Outcome/<br>Study Drug Action Taken/ Serious?/<br>Other Action Taken Criteria M | Serious?/<br>Criteria Met | TEAE?<br>[2] |
|---|---|---|---|---|---|---|---|
| XXXX | XXXXXX | XXXXXXXXXXX/<br>XXXXXXXXXXXXXXXXXXXXXXXXX | DDMMMYYYY/hh:mm (X)/<br>DDMMMYYYY/hh:mm (X) | XXXXXXXXXX | ************************************** | × | × |
| XXXX | XXXXXXX | Xxxxxxxxxxx/<br>Xxxxxxxxxxx/<br>Xxxxxxxxxxxxx | DDMMMYYYY/hh:mm (X)/<br>DDMMMYYYY/hh:mm (X) | /XXXXXXXXX | ************************************** | × | × |

Abbreviations: TEAE = Treatment emergent adverse event.

Note: Study day is calculated relative to the date of first dose of study drug. AEs were coded using MedDRA version 20.1

[1] Treatment groups are based on treatment received. The dose received at the beginning of the treatment-phase, or the last dose received if the subject discontinued from the study during the treatment-phase, is presented. \* = subject was down-titrated due to tolerability issues.

[2] A TEAE is any AE with an onset date/time between the initiation of study drug and 5 days after the last dose of study drug. This will include any AE with onset prior to initiation of study drug and increased severity after the treatment administration.

SOURCE: Listing 16.2.7.1

Programming note: If time missing, display "----". "Other Action Taken" will be either None, Concomitant Medication, Non-drug Therapy, or Other; if specify text is needed, concatenate "Concomitant Medication:" or "Other:" with the text. If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. If no events meet the criteria for display, present "No events are reported." SOC & PT text should be in proper case in table, as shown in the shell. TEAE will be Yes or No. Since treatment groups presented are based on the dose (mg) received at the beginning of the treatment-phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to to the source in the column. Add "16.2.5.2" to the SOURCE line.



Table 14.3.3.1.2 Listing of Adverse Events Leading to Study Drug Discontinuation Dose-Optimization Safety Population

#### (Same shell as Table 14.3.3.1.1)

Programming Note: Update footnote [1] to read "Treatment groups are based on treatment received. The optimized dose is presented."





Table 14.3.3.2.1 Listing of Serious Adverse Events Treatment-Phase Safety Population

(Same shell as Table 14.3.3.1.1)

Table 14.3.3.2.2 Listing of Serious Adverse Events Dose-Optimization Safety Population

(Same shell as Table 14.3.3.1.1)

Programming Note: Update footnote [1] to read "Treatment groups are based on treatment received. The optimized dose is presented."



**premier** research



(Same shell as Table 14.3.3.1.1)

Table 14.3.3.2 Listing of Deaths Dose-Optimization Safety Population

(Same shell as Table 14.3.3.1.1)

Programming Note: Update footnote [1] to read "Treatment groups are based on treatment received. The optimized dose is presented."



Table 14.3.3.4.1 Incidence of Abuse Related Adverse Events by SOC, PT, and Treatment Treatment-Phase Safety Population

| | | KP415 | | | |
|---|---|---|---|---|---|
| System Organ Class | 20 mg<br>(N=XX) | 30 mg<br>(N=XX) | 40 mg<br>(N=XX) | δ̈̈́, | Overall (N=XX) |
| Preferred Term | , n (%) | n (%) n | , (%) n | u (%) | , 95% CI |
| Subjects with at least 1 Abuse<br>Related TEAE | XX (XX.X%) | XX (XX.X%) | (%X:X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| System Organ Class 1 | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Preferred Term 1 | (%X:XX) XX | (%X:X%)<br>XX | (%X:XX) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Preferred Term 2 | (%X:XX) XX | (%X:X%) | (%X:XX) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Preferred Term 3 | (%X:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| System Organ Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Preferred Term 1 | (%X:XX) XX | (%X:X%) | (%X:XX) XX | (XX:X%) | (XX.X%, XX.X%) |
| Preferred Term 2 | (%X:XX) XX | (%X:X%)<br>XX | (%X:XX) XX | (XX:X%) | (XX.X%, XX.X%) |
| Preferred Term 3 | (%X:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |

beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. AEs were coded using MedDRA Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Treatment groups are based on treatment received. The dose received at the Abbreviations: CI = confidence interval; PT = Preferred Term; SOC = System Organ Class.

version 20.1. AEs that are abuse potential-related include the following MedDRA PTs: euphoria-related terms, terms of altered attention, cognition and mood, and dissociative/psychotic terms. A treatment related TEAE is an AE that is marked as being possibly, probably, or definitely related to treatment. Subjects are counted once for each SOC and once for each PT. AEs are displayed by descending frequency of SOC, then PT within SOC, and then alphabetically by PT. 95% Wilson CIs are presented.

SOURCE: Listing 16.2.7.1

Programming note: SOC & PT text should be in proper case in table, as shown in the shell. Ensure correct MedDRA version is printed in footnote. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add "16.2.7 to the SOURCE line.



Incidence of Abuse Related Adverse Events by SOC, PT, and Age Treatment-Phase Safety Population Table 14.3.3.4.2

#### (Same shell as Table 14.3.3.4.1)

Programming note: Column headers will be "Overall", and each appropriate Age range. Check cut points per Section 9.1.3 of SAP. Remove footnote explaining treatment groups.

Table 14.3.3.4.3 Incidence of Abuse Related Adverse Events by SOC, PT, and Gender Treatment-Phase Safety Population

#### (Same shell as Table 14.3.3.4.1)

Programming note: Column headers will be "Overall", "Male", and "Female." Remove footnote explaining treatment groups.

Table 14.3.3.4.4 Incidence of Abuse Related Adverse Events by SOC, PT, and Treatment Dose-Optimization Safety Population

#### (Same shell as Table 14.3.3.4.1)

Programming Note: Update footnote to read "Treatment groups are based on treatment received. The optimized dose is presented."




Table 14.3.5.1.1 Summary of Hematology Laboratory Results by Study Visit and Treatment Treatment-Phase Safety Population

Parameter: XXXXXXXXX

| | x) all | CFB | | | | | × | XX.X (XX.XX) | XX.XX | ×:× | ×,× | } | <b>\( \)</b> | XX.XX)<br>XX.XX) | XX.XX | ××× | ××× |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Overall (N=XX) | Observed | × | (XX.XX)<br>XX.XX | XXX | X, X | | XX.X (XX.XX) | | | | | | | | | ×<br>×<br>× |
| | mg<br>XX) | CFB | | | | | × | XX.X (XX.XX) | XX.X | ×:× | ××× | } | <b>\{</b> | XX:XX) | XX.XX | ××× | ××× |
| | 40 mg<br>(N=XX) | Observed | × | (XX XX)<br>X X X X X X X X X X X X X X X X X | XXX | ××× | × | XX.X (XX.XX) | XX.X | ××× | X<br>X<br>X | } | <b>\(\)</b> | XX.XX) X.XX | XX:XX | ××× | ××× |
| 15 | mg<br>XX) | CFB | | | | | × | XX.X (XX.XX) | XX.XX | ××× | ××× | } | <del>×</del> | XX.XX) X.XX | XX.XX | ××× | ××× |
| KP415 | 30 mg<br>(N=XX) | Observed | × | (XX XX)<br>X X X X X X X X X X X X X X X X X | XX | ××× | × | XX.X (XX.XX) | XX.XX | ×:× | XX<br>XX | } | <b>\{</b> | XX.XX) X.XX | XX:XX | ×.× | ××× |
| | gr<br>(X | CFB | | | | | × | XX.X (XX.XX) | XX.XX | ××× | ×,× | } | <b>\{</b> | XX.XX) | XX:XX | ×:× | ××× |
| | 20 mg<br>(N=XX) | Observed | × | (XX:XX)<br>XX:XX<br>XX:XX | XXX | XX, XX | × | XX.X (XX.XX) | ××:×× | X:X | ××× | } | <del>\</del> | (XX:XX) | ××:×× | X:X | ×× |
| | Study Visit | Statistic | Baseline [1]<br>n | Mean (SD)<br>CV% | Median | Min, Max | Visit 11<br>n | Mean (SD) | %\C | Median | Min, Max | Visit 17 | = | Mean (SD) | %\C | Median | Min, Max |

## Continue for other parameters. Sort alphabetically by parameter.

Abbreviations: CFB = change from baseline. CV% = coefficient of variation; NA = not applicable; SD = standard deviation.

Note: Treatment groups are based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from

the study during the Treatment Phase, is presented.
[1] Baseline is the Screening Visit 01A for new subjects and either the Screening Visit 01B or the last KP415.E01 Study Visit for roll-over subjects. SOURCE: Listing 16.2.8.1.1

Programming note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add "16.2.5.2" to the SOURCE line.



Shift from Baseline in Hematology Laboratory Results by Study Visit and Treatment Treatment-Phase Safety Population Table 14.3.5.1.2

Parameter: XXXXXXX

| | | Baseline [1] | le [1] | |
|---|---|---|---|---|
| | | KP415 Overall (N=XX | all (N=XX) | |
| Study Visit | Low | Normal | High | Missing |
| Category | n (%) | n (%) | n (%) | n (%) |
| Visit 11 | | | | |
| Low | XX (XX:X%) | (XX:X%) | XX (XX: X%) | (%X:X%) |
| Normal | (%X:XX) | XX (XX: X%) | (%X:XX) XX | XX (XX:X%) |
| High | (%X:XX) | (%X:XX)<br>XX | (%X:XX)<br>XX | (%X:XX) XX |
| Missing | (%X:XX) | (%X:XX)<br>XX | (%X:XX)<br>XX | (%X:XX)<br>XX |
| | | | ( | |
| Visit 17 | | | | |
| Low | XX (XX:X%) | (%X:X%) | XX (XX: X%) | (%X:X%) |
| Normal | (%X:X%) | (%X:X%) XX | (%X.XX) XX | (%X:XX) XX |
| High | XX (XX: X%) | (%X:X%) XX | (%X:X%) | (%X:XX) XX |
| Missing | XX (XX.X%) | XX (XX.X%) | XX (XX: X%) | XX (XX.X%) |

# Continue for other parameters and treatment groups. Sort alphabetically by parameter.

Abbreviations: CFB = change from baseline; NA = not applicable.

by treatment received. Treatment groups are based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented.
[1] Baseline is the Screening Visit 01A for new subjects and either the Screening Visit 01B or the last KP415.E01 Study Visit for roll-Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Subjects are summarized overall and

over subjects. SOURCE: Listing 16.2.8.1.1

Programming note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment-Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject receives a lower dose than planned due to tolerability issues."; add "16.2.5.2" to the SOURCE line.



Summary of Serum Chemistry Laboratory Results by Study Visit and Treatment Treatment-Phase Safety Population Table 14.3.5.2.1

(Same shell as Table 14.3.5.1.1; SOURCE: Listing 16.2.8.1.2)

Table 14.3.5.2.2 Shift from Baseline in Serum Chemistry Laboratory Results by Study Visit and Treatment Treatment-Phase Safety Population

(Same shell as Table 14.3.5.1.2; SOURCE: Listing 16.2.8.1.2)

Table 14.3.5.3.1 Summary of Quantitative Urinalysis Laboratory Results by Study Visit and Treatment Treatment-Phase Safety Population

(Same shell as Table 14.3.5.1.1; SOURCE: Listing 16.2.8.1.3)

Table 14.3.5.3.2 Shift from Baseline in Quantitative Urinalysis Laboratory Results by Study Visit and Treatment Treatment-Phase Safety Population

(Same shell as Table 14.3.5.1.2; SOURCE: Listing 16.2.8.1.3)



Table 14.3.5.3.3 Summary of Qualitative Urinalysis Laboratory Results by Study Visit and Treatment Treatment-Phase Safety Population

Parameter: XXXXXXXX

| | | KP415 | | | |
|---|---|---|---|---|---|
| Study Visit | 20 mg<br>(N=XX) | 30 mg<br>(N=XX) | 40 mg<br>(N=XX) | δŻ | Overall (N=XX) |
| Category | n (%) <sup>(</sup> | , (%) u | n (%) | u (%) | , 95% CI |
| Baseline [1]<br>Category 1 | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX:X%, XX:X%) |
| Category 2<br>Category 3 | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | (XX.X%, XX.X%)<br>(XX.X%, XX.X%) |
| Visit 11<br>Category 1 | XX (XX.X%) | XX (XX.X%) | (%X:X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Category 2<br>Category 3 | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | (XX.X%, XX.X%)<br>(XX.X%, XX.X%) |
| Visit 17<br>Category 1 | (%X:XX) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Category 2<br>Category 3 | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | (XX.X%, XX.X%)<br>(XX.X%, XX.X%) |

Continue for other parameters. Sort alphabetically by parameter.

Abbreviation: CI = confidence interval; NA = not applicable.

based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. 95% Wilson Cls are presented. Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Subjects are summarized overall and by treatment received. Treatment groups are

[1] Baseline is the Screening Visit 01A for new subjects and either the Screening Visit 01B or the last KP415.E01 Study Visit for roll-over subjects. SOURCE: Listing 16.2.8.1.3

Programming note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment-Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add "16.2.5.2" to the SOURCE line.





Table 14.3.6.1 Summary of Vital Signs by Study Visit and Treatment Treatment-Phase Safety Population (Same shell as Table 14.3.5.1.1; visits include Baseline, Visit 3 and Visit 4 for new subjects in the Dose Optimization Phase, Visit 5-Visit 17 for subjects in the Treatment-Phase; parameters include Temperature (C), pulse Rate (bpm), Respiratory Rate (breaths per min) Sitting Systolic Blood Pressure (mmHg), Height (cm), and Weight (kg), BMI (kg/m²); ensure footnote updated to SOURCE: Listing 16.2.8.2)

Table 14.3.6.2.1 Summary of 12-Lead Electrocardiogram by Study Visit and Treatment Treatment-Phase Safety Population (Same shell as Table 14.3.5.1.1; visits include Baseline, Visit 3 and Visit 4 for new subjects in the Dose Optimization Phase, Visit 5-Visit 17 for subjects in the Treatment-Phase; parameters include HR, RR, QT, QTcF; ensure footnote updated to SOURCE: Listing 16.2.8.3)



Summary of 12-Lead Electrocardiogram Interpretation by Study Visit and Treatment Treatment-Phase Safety Population Table 14.3.6.2.2

| | | KP415 | | | |
|---|---|---|---|---|---|
| Study Visit | 20 mg<br>(N=XX) | 30 mg<br>(N=XX) | 40 mg<br>(N=XX) | ô <sup>'</sup> | Overall (N=XX) |
| Category | (%) u | u (%) | u (%) | u (%) | 95% CI |
| Baseline [1]<br>Nomal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | (XX.X%, XX.X%)<br>(XX.X%, XX.X%) |
| Visit 11<br>Nomal | XX (XX.X%) | XX (XX.X%) | (%X:XX) | XX (XX.X%) | (XX.X%, XX.X%) |
| Abnormal, Not Clinically Significant<br>Abnormal, Clinically Significant | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | XX (XX.X%)<br>XX (XX.X%) | (XX.X%, XX.X%)<br>(XX.X%, XX.X%) |
| Visit 17<br>Nomal | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX:X%, XX:X%) |
| Abnormal, Not Clinically Significant | (%X:X%)<br>XX | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Abnormal, Clinically Significant | (%X:X%) | XX (XX:X%) | XX (XX.X%) | XX (XX:X%) | (XX:X%, XX:X%) |

Abbreviation: CI = confidence interval; NA = not applicable.

Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Treatment groups are based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. 95% Wilson CIs are presented. [1] Baseline is the Screening Visit 01A for new subjects and either the Screening Visit 01B or the last KP415.E01 Study Visit for roll-over subjects. SOURCE: Listing 16.2.8.3 Programming note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment-Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add "16.2.5.2" to the SOURCE line.



Summary of Columbia-Suicide Severity Rating Scale (C-SSRS) Treatment-Phase Safety Population Table 14.3.6.3

| | | KP | KP415 | |
|---|---|---|---|---|
| | 20 | 20 mg | 30 | 30 mg |
| C-SSRS Section | Pre-treatment | Post-treatment | Pre-treatment | Post-treatment |
| C-SSRS Item | (N=xx) | (N=XX) | (N=xx) | (N=xx) |
| : | | | | |
| Suicidal Ideation | (%X:XX) XX | (%X:XX)<br>XX | (%X:XX)<br>XX | (%X:X%)<br>XX |
| Wish to be Dead | (%X:XX) XX | (%X:X%) | (%X:XX) XX | (%X:X%) |
| Non-Specific Active Suicidal Thoughts | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (%X:X%) XX |
| Active Suicidal Ideation with Any Methods | XX (XX.X%) | (%X:X%) | (%X:XX) XX | (%X:X%) XX |
| Active Suicidal Ideation with Some Intent | XX (XX.X%) | XX (XX: X%) | (%X:XX) XX | (XX.X%) |
| Active Suicidal Ideation with Specific Plan | XX (XX.X%) | XX (XX.X%) | (%X:X%) | XX (XX.X%) |
| Suicidal Behavior | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Actual Attempt | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (%X:X%) XX |
| Subject Engaged in Non-Suicidal Self- | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Injurious Behavior | | | | |
| Interrupted Attempt | (%X:X%) | (%X:X%) | (%X:XX) XX | (%X:X%) |
| Aborted Attempt | (%X:XX) XX | XX (XX: X%) | (%X:XX) | (%X:X%) |
| Preparatory Acts or Behavior | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX |
| Suicidal Behavior | XX (XX.X%) | (%X:XX) XX | (%X:XX) XX | (%X:X%) XX |
| Suicide | XX (XX.X%) | (%X:XX) XX | (%X:X%) | XX (XX.X%) |

during the Treatment Phase, is presented. The C-SSRS scale consists of a Screening evaluation that assesses the lifetime and more recent experience (past 6 months) of the subject with suicidal ideation and behavior, a baseline evaluation that focuses on suicidality since received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study ("post-treatment") that focuses on suicidality since the last study visit. Subjects are counted once for each C-SSRS section and once for each C-SSRS item answered "Yes" in pre-treatment and post-treatment. Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Treatment groups are based on treatment Screening that occurs before first dose of study drug (all of which is summarized under "pre-treatment"), and a post-baseline evaluation

SOURCE: Listing 16.2.8.4

Programming note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add data. If a subject receives a lower dose than planned due to tolerability, this SOURCE line.

AD-ST-33.05 Effective date: 22-Jan-2018

Version 0.1 | 07-Jun-2018 | AD-PR-109.01 Effective date: 26-Jun-2017



| | Treatment-Phase | Treatment-Phase Safety Population | | |
|---|---|---|---|---|
| | Α | KP415 | | |
| | 40 | 40 mg | Ŏ | Overall |
| S Section | Pre-treatment | Post-treatment | Pre-treatment | Post-treat |
| RS Item | (x=x) | (N=xx) | (N=xx) | (N=xx |
| l Ideation | XX (XX:X%) | XX (XX.X%) | XX (XX.X%) | (XX) XX |
| to be Dead | XX (XX:X%) | XX (XX.X%) | (%X:XX) XX | (XX)<br>XX |

| | 40 | 40 mg | ŏ | Overall |
|---|---|---|---|---|
| C-SSRS Section | Pre-treatment | Post-treatment | Pre-treatment | Post-treatment |
| C-SSRS Item | (N=xx) | (N=xx) | (N=xx) | (N=xx) |
| Suicidal Ideation | (%X:X%) XX | (%X:XX) | (%X:XX) | (%X:X%) |
| Wish to be Dead | XX (XX:X%) | (%X:X%)<br>XX | (%X:XX) | (%X:XX) XX |
| Non-Specific Active Suicidal Thoughts | (%X:X%) | (%X:XX) XX | (%X:XX) | (%X:X%) XX |
| Active Suicidal Ideation with Any Methods | (%X:X%) | (%X:X%) XX | (%X:XX) | XX (XX:X%) |
| Active Suicidal Ideation with Some Intent | (XX:X%) | (%X:XX) XX | (%X:XX) | (%X:XX) XX |
| Active Suicidal Ideation with Specific Plan | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Suicidal Behavior | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Actual Attempt | XX (XX:X%) | (XX:X%) | (%X:XX) | XX (XX.X%) |
| Subject Engaged in Non-Suicidal Self-<br>Iniurious Behavior | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) |
| Interrupted Attempt | XX (XX:X%) | XX (XX.X%) | XX (XX:X%) | XX (XX.X%) |
| Aborted Attempt | XX (XX:X%) | XX (XX.X%) | (%X:XX) | XX (XX.X%) |
| Preparatory Acts or Behavior | XX (XX:X%) | (XX:X%) | (%X:XX) XX | (%X:XX) XX |
| Suicidal Behavior | XX (XX:X%) | (%X:X%) XX | (%X:XX) XX | (%X:XX) XX |
| Suicide | (%X:X%) XX | (%X.XX) | (%X:X%) | (%X:XX) XX |

during the Treatment Phase, is presented. The C-SSRS scale consists of a Screening evaluation that assesses the lifetime and more recent experience (past 6 months) of the subject with suicidal ideation and behavior, a baseline evaluation that focuses on suicidality since received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study ("post-treatment") that focuses on suicidality since the last study visit. Subjects are counted once for each C-SSRS section and once for each C-SSRS item answered "Yes" in pre-treatment and post-treatment. Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Treatment groups are based on treatment Screening that occurs before first dose of study drug (all of which is summarized under "pre-treatment"), and a post-baseline evaluation

SOURCE: Listing 16.2.8.4

Programming note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add "16.2.5.2" to the SOURCE line.



Summary of Concomitant Medications by ATC Class Level 4, PT, and Treatment Treatment-Phase Safety Population Table 14.3.6.4

| | | KP415 | | | |
|---|---|---|---|---|---|
| ATC Class Level 4 | 20 mg<br>(N=XX) | 30 mg<br>(N=XX) | 40 mg<br>(N=XX) | ÒZ. | Overall (N=XX) |
| Preferred Term (ATC Class Level 5) | n (%) | u (%) | n (%) | u (%) | 95% CI |
| Subjects with at least 1 Concomitant<br>Medication | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| ATC Class 1 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Preferred Term 1 | (%X:X%) XX | (%X:XX) XX | (%X:XX) XX | (%X:X%) | (XX.X%, XX.X%) |
| Preferred Term 2 | (%X:X%) XX | (%X:XX) XX | (%X:XX) XX | (XX.XX) | (XX.X%, XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| ATC Class 2 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |
| Preferred Term 1 | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Preferred Term 2 | (%X:X%) XX | (%X:XX) XX | (%X:XX) XX | (%X:XX) XX | (XX.X%, XX.X%) |
| Preferred Term 3 | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | (XX.X%, XX.X%) |

Abbreviations: ATC = Anatomical Therapeutic Chemical; CI = confidence interval; PT = Preferred Term.

Note: Percentages are n/Number of subjects in the Treatment-Phase Safety Population\*100. Treatment groups are based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. 85% Wilson Cisare presented. Medications were coded using WHO-DDE version September 2017. Concomitant medications are all medications that were continuing or starting after first dose of study drug. Medications are displayed by descending frequency of Anatomic Therapeutic Chemical (ATC) Level 4 classification, by PT within ATC, and then alphabetically. Subjects were counted only once for each ATC and PT. 95% Wilson CIs are presented. SOURCE: Listing 16.2.8.6

based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, this should be mentioned in the footnote as "Subject XXXXXX was down-titrated due to tolerability issues."; add "16.2.5.2" to the SOURCE line. Programming note: ATC & PT text should be in proper case in table, as shown in the shell. Ensure correct WHO-DDE is printed in footnote. Since treatment groups presented are



Planned Listing Shells

13.9.



**premier** research



Listing 16.2.1 Subject Disposition All Subjects

| Subject ID | Subject ID Treatment [1] | Site | Did Subject<br>Complete<br>Study? | Date of Completion/Discontinuation (Study Day) | Date of Last Visit<br>(Study Day) | Reason for Discontinuation | Last Dose Received Prior to Discontinuation |
|---|---|---|---|---|---|---|---|
| XXXXXX | XXXXXX | XXXXXX | Yes | DDMMMYYYY (XX) | DDMMMYYYY (XX) | | |
| XXXXXX | XXXXXX | XXXXX | Yes | DDMMMYYYY (XX) | DDMMMYYYY (XX) | | |
| XXXXXX | XXXXXX | XXXXX | Yes | DDMMMYYYY (XX) | DDMMMYYYY (XX) | | |
| XXXXXX | XXXXXX | XXXXX | N<br>N | DDMMMYYYY (X) | DDMMMYYYY (X) | XXXXXXXX: XXXXXXXX | XXX |
| XXXXXX | XXXXXX | XXXXXX | o<br>N | DDMMMYYYY (XX) | DDMMMYYYY (XX) | DDMMMYYYY (XX) XXXXXXXXXXXXXXXXXXXX | XXX |

Abbreviation: NA = not applicable.

Note: Study day is calculated relative to the date of first dose of study drug.
[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* subject was down-titrated due to tolerability issues.

concatenate with date of last contact as follows: "Lost to follow-up; date of last contact: DDMMMYYYY". Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the Programming Note: If reason for early termination is Other, concatenate the specify text as follows: "Other: XXXXXXXXX". If reason for early termination is lost to follow-up,

treatment in the treatment column.



Listing 16.2.2.1 Inclusion and Exclusion Criteria Not Met All Subjects

| Any Exclusion<br>Criteria Met? | [3] | o<br>N | o<br>N | o<br>N | Yes: 05 | o<br>N | oN<br>N |
|---|---|---|---|---|---|---|---|
| All Inclusion<br>Criteria Met? | [2] | Yes | No: 02, 07 | No: 02 | Yes | Yes | Yes |
| Day) of: | Informed Assent | DDMMMYYYY (-X) | ррмммүүүү (-X) | ррмммүүүү (-X) | ррмммүүүү (-X) | ррмммүүүү (-X) | DDMMMYYYY (-X) |
| Date (Study Day) of: | Screening/Informed Consent | DDMMMYYYY (-X) | DDMMMYYYY (-X) | DDMMMYYYY (-X) | DDMMMYYYY (-X) | DDMMMYYYY (-X) | DDMMMYYYY (-X) |
| | Subject ID Treatment [1] | XXXXXX | ××××× | ××××× | ××××× | ××××× | XXXXXX |
| | Subject ID | XXXXXX | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |

Note: Study day is calculated relative to the date of first dose of study drug.

Disorders - Fifth Edition (DSM-5) criteria for a primary diagnosis of ADHD (combined, inattentive, or hyperactive/impulsive presentation) per clinical evaluation and confirmed by the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID). If the MINI-KID 2] 02 Subject must have a body weight of at least 21 kg at Screening: 07 = Subject must meet Diagnostic and Statistical Manual of Mental 1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues. assessment is available from a previous study with KP415, it does not need to be repeated.

[3] 05 = Subject has a positive urine MPH screen at Visit 5.

in the example. If no criteria are present for a column, remove the [2] and/or [3] from the column header. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment-Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the Programming note: If more than 1 inclusion or exclusion criterion number exists, concatenate with a comma as shown above. Decode any relevant criteria in the footnotes as shown treatment in the treatment column. **premier** research



| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | MAJOR | XXXXXXXXXXX | XXXXXXXX | XXXXX |
|---|---|---|---|---|
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | MINOR | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXX | XXXXX |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | MAJOR<br>MINOR | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXX | XXXXX |
| Description | Violation<br>Level | Event Type | Subject ID Treatment [1] | Subject ID |

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

Programming note: The structure of this listing may change depending on the information in the protocol deviations file. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to treatment in the treatment column.



Listing 16.2.3 Analysis Populations All Subjects

| l | ĺ | | | |
|---|---|---|---|---|
| | Reason(s) for Exclusion | Dose-Optimization Safety Population:<br>Subject did not have at least 1 post-dose<br>safety assessment in the Dose<br>Optimization Phase. | | Treatment-Phase Safety: Subject did not receive at least 1 dose of study drug. |
| Dose-<br>Optimization | Safety<br>[4] | o<br>N | Yes | o<br>Z |
| | Efficacy<br>[3] | Yes | Yes | <u>8</u> |
| Treatment-<br>Phase | Safety<br>[2] | Yes | Yes | 8<br>N |
| | Subject ID Treatment [1] | XXXXX | XXXXXXX | XXXXX |
| | Subject ID | XXXXXX | XXXXXX | XXXXX |

Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the Programming note: Concatenate all reasons for exclusion with a semi-colon. Since treatment groups presented are based on the dose (mg) received at the beginning of the treatment column.

<sup>[1]</sup> Treatment is based on treatment received. The dose received at the beginning of the treatment-phase, or the last dose received if the subject discontinued from the study during the treatment-phase, is presented. [2] The Treatment-Phase Safety Population includes all subjects who are enrolled in the Treatment Phase and

received at least 1 dose of study medication in the Treatment Phase and had at least 1 post-dose safety assessment in the Treatment Phase. \* = subject was down-titrated due to tolerability issues.

Treatment Phase and had adequate data to assess the change from baseline of the efficacy parameters and who [3] The Efficacy Population includes all enrolled subjects who received at least 30 days of study medication in the had no protocol deviations that could affect the efficacy parameters.

<sup>[4]</sup> The Dose-Optimization Safety Population includes all subjects who are enrolled in the Dose Optimization Phase and received at least 1 dose of study medication in the Dose Optimization Phase and had at least 1 post-dose safety assessment in the Dose Optimization Phase.



Listing 16.2.4.1 Demographics and Baseline Characteristics All Subjects

| Subject ID | Subject ID Treatment [1] | Sex | Child-Bearing<br>Potential? | Date of<br>Birth | Age<br>(years) | Ethnicity | Race | Weight<br>(kg) | Height<br>(cm) | BMI<br>(kg/m²) | BSA $(m^2)$ [2] |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXXXXX | XXXX | XXXX | | DDMMMYYY | × | XXXXXXX | XXXXXXX | X:X | ×× | XX.XX | XX.XX |
| XXXXX | XXXXXX | XXXXXX | N <sub>o</sub> | DDMMMYYY | × | XXXXXXX | XXXXX | ×× | × | XX.XX | XX.XX |
| XXXXX | XXXXXX | XXXXXX | Yes | DDMMMYYY | × | XXXXXXX | XXXXX | ×× | × | XX.XX | XX.XX |
| XXXXX | XXXX | ××× | | DDMMMYYY | × | XXXXXXX | XXXX | ×× | × | XX.XX | XX.XX |
| XXXXX | XXXXXX | XXXXXX | Š | DDMMMYYY | × | XXXXXXX | XXXXX | ×× | × | XX.XX | XX.XX |
| XXXXXX | XX | XXXX | | DDMMMYYY | × | XXXXXX | XXXXXX | ××× | ××× | XX.XX | XX.XX |

Programming Note: If race is other, concatenate "Other:" with specify text. If subject has multiple races, concatenate them. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment column.

Abbreviation: BMI = Body Mass Index; BSA = body surface area.

Note: Height, weight, BMI, and BSA are the values at Screening.

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

<sup>[2]</sup> BSA = $\sqrt{[\text{height(cm)} * \text{weight(kg)}]/3600}$ 



**premier** research

Listing 16.2.4.2 Medical History All Subjects

| Start Date (Study Day)/<br>End Date (Study Day)/ | DDMMMYYYY (X)/<br>DDMMMYYYYY (X) | MIMMYYYY (X)/<br>Ongoing | MIMMYYYY (X)/<br>Ongoing | DDMMMYYYY $(X)/$ DDMMMYYYY $(X)$ |
|---|---|---|---|---|
| System Organ Class/<br>Preferred Term/<br>Verbatim Term | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | /xxxxxxxxxx/<br>/xxxxxxxxxxxxxxxxxxxxxxxx | /xxxxxxxxxx/<br>/xxxxxxxxxxxxxxxxxxxxxxxx | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Treatment [1] | XXXXXXXX | | | XXXXXXXX |
| Subject ID | XXXXX | | | XXXXX |

Note: Study day is calculated relative to the date of first dose of study drug. Medical history was coded using MedDRA version 20.1. Only subjects with medical history recorded are listed.
[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

Programming note: SOC & PT text should be in proper case in table, as shown in the shell. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column.



Listing 16.2.4.3 ADHD Diagnosis and Confirmation All Subjects

| Date of ADHD Diagnosis<br>(Study Day) | DDMMMYYYY (X) | DDMMMYYYY (X) |
|---|---|---|
| Subject ID Treatment [1] Has an ADHD Diagnosis been confirmed? | XXX | XXX |
| Treatment [1] | XXXXXXXX | XXXXXXXX |
| Subject ID | XXXXXX | XXXXXX |

Abbreviations: ADHD = attention-deficit hyperactivity disorder Note: Study drug.

Note: Study day is calculated relative to the date of first dose of study drug.

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability

Programming note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column.



Listing 16.2.4.4 Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) All Subjects

| | | Was | | Interview | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Treatment<br>[1] | Treatment Assessment [1] Performed? | Date (Study<br>Day) | Start/Stop<br>Time | Total Time | Module | ltem | Response | Primary Diagnosis? |
| XXXXXX | XXXXX | XXXX | DDMMMYYYY<br>(-x) | hh:mm/ | XXXX | Major Depressive<br>Enisode | Current (Past 2 weeks) | × | |
| | | | (***) | | | | Past | × | |
| | | | | | | | Recurrent | × | |
| | | | | | | Major Depressive | Current (Past 2 weeks) | × | XXX |
| | | | | | | Disorder | | | |
| | | | | | | | Past | × | ××× |
| | | | | | | | Recurrent | × | ××× |
| | | | | | | Suicidality | Current (Past Month) | × | XXX |
| | | | | | | • | Lifetime | × | ××× |
| | | | | | | | Lifetime Attempt Level | XXXXX | |
| | | | | | | | | × | |
| | | | | | | Suicide Behavior<br>Disorder | Current (In Past Year) | × | XXX |
| | | | | | | | In early remission (1-2 years ago) | × | XXX |
| | | | | | | : | | | |

Abbreviations: MINI-KID= Mini International Neuropsychiatric Interview for Children and Adolescents
[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

Programming note: Continue for other categories and assessments. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column. 



**premier** research



| XXXXXXX XXXXXXX | |
|-----------------|-----|
| | XXX |
| XXXXXXX | XXX |
| XXXXXXX XXXXXX | XXX |
| xxxxxx | XXX |

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

Programming note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to treatment in the treatment column.



Listing 16.2.5.2 Study Drug Dispensation and Return All Subjects

| Subject<br>Compliant?<br>(% Compliance)<br>[2] | Yes (100%) | | Yes (80%) | | No (60%): | *************************************** | Yes (100%) | | Yes (85%) |
|---|---|---|---|---|---|---|---|---|---|
| Number of Doses<br>Missed (Reason) | × | | (XXXX) XX | | (XXXX) XX | | × | | (XXXX) XX |
| Adjusted<br>Dose<br>Level (mg) | × | × | | × | | × | | × | |
| Dose<br>Adjusted? | o<br>Z | Š | | Yes: XXXX | | <sub>S</sub> | | <sub>o</sub> | |
| Number of<br>Capsules<br>Dispensed/<br>Returned | ×× | × | × | × | × | × | × | × | × |
| Date Dispensed/<br>Returned<br>(Study Day) | DDMMMYYYY (X)<br>DDMMMYYYY (X) | DDMMMYYYY (XX) | DDMMYYYY (XX) | DDMMYYYY (XX) | DDMMMYYYY (XX) | DDMMMYYYY (XX) | DDMMMYYYY (XX) | DDMMMYYYY (X) | DDMMMYYYY (X) |
| Study<br>Medication<br>Dispensed/<br>Returned? | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| Study<br>Medication<br>Assessment<br>Type | Dispensed<br>Returned | Dispensed | Returned | Dispensed | Returned | Dispensed | Returned | Dispensed | Returned |
| Study Visit | Visit 2 | Visit 3 | | Visit 4 | | Visit 5 | | Visit 6 | |
| Subject ID Treatment [1] | ××××××× ×××××× | | | | | | | | |
| Subject ID | XXXXX | | | | | | | | |

Note: Study day is calculated relative to the date of first dose of study drug.
[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the

Programming note: If med not dispensed or returned, or subject is not compliant, concatenate reason like: "No: XXXXXX". If Dose was adjusted, concatenate reason like: "He XXXXXX". If Any doses were missed, concatenate reason like: "#: XXXXXX".

Treatment Phase, is presented. [2] Acceptable compliance is defined as 80-100% of total doses (inclusive).



Listing 16.2.6.1 ADHD-Rating Scale-5 All Subjects

| Text Result | XXXXXXXX | XXXXXXXX | XXXXXXX | XXXXXXX | XXXXXXX | | |
|---|---|---|---|---|---|---|---|
| Numeric<br>Result | × | × | × | × | × | × | × × |
| Assessment | Fails to give close attention to details or XX makes careless mistakes in schoolwork or during other activities | Has difficulty sustaining attention in tasks or play activities | Does not seem to listen when spoken to directly | Does not follow through on instructions and fails to finish schoolwork or chores | Has difficulty organizing tasks and activities | Inattention Subscale Score | Hyperactivity/Impulsivity Subscale<br>Score<br>Total ADHD-RS-5 Score |
| Category | How often does your<br>child display this<br>behavior? | | | | | Subscale and Total Scores | |
| Date of Assessment<br>(Study Day) | XXXXXX XXXXXX DDMMMYYYY (XX) | | | | | | |
| Study<br>Visit | × | | | | | | |
| Subject Treatment Study<br>ID [1] Visit | ×××× | | | | | | |
| Subject<br>ID | XX-XXX | | | | | | |

Note: Study day is calculated relative to the date of first dose of study drug.

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment-Phase, is presented. \* = subject was down-titrated due to tolerability issues.

[2] Change from baseline is calculated as Numeric Result – Baseline.

Programming Note: Continued for other categories and assessments. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment

AD-ST-33.05 Effective date: 22-Jan-2018

Version 0.1 | 07-Jun-2018 | AD-PR-109.01 Effective date: 26-Jun-2017



Listing 16.2.6.2 Clinical Global Impression (CGI) – Severity All Subjects

| | Text | Result | XXXXXX | XXXXXX |
|---------|------------|---------------|---------------|---------------|
| | Numeric | Result | × | × |
| | Reason Not | Performed | | |
| Date of | Assessment | (Study Day) | DDMMMYYYY (X) | DDMMMYYYY (X) |
| | | ] Study Visit | XXXXXX | XXXXXXX |
| | | Treatment [1] | XXXXXX | |
| | Subject | ₽ | XX-XX | |

Abbreviation: CGI-S = Clinical Global Impression - Severity.

Note: Study day is calculated relative to the date of first dose of study drug. The CGI-S score is based on the following question regarding severity of illness: Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues. Programming note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column.



**premier** research

Listing 16.2.6.3 Clinical Global Impression (CGI) – Improvement All Subjects

### Same shell as Listing 16.2.6.2; use the following footnotes:

Abbreviation: CGI-I = Clinical Global Impression – Improvement.

Note: Study day is calculated relative to the date of first dose of study drug. The CGI-I score is based on the following question regarding global improvement: Rate total improvement whether or not, in your judgment, it is due entirely to drug treatment. Compared to his/her condition at admission to the project, how much has patient changed?



Listing 16.2.6.4 Children's Sleep Habits Questionnaire (CSHQ) All Subjects

| Text Result | hh:mm | XXXXXX | XXXXXXXX | XXXXXXXX | XXXXX | XXXXXXX | XXXXXXXX | | XXXXX | XXXXXXXX | XXXXX | XXXXXXX | XXXXXXXX | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Numeric<br>Result | | × | × | × | × | × | × | | × | × | × | × | × | × | × | × | × |
| Assessment | Child's bedtime | <ol> <li>Child goes to bed at the same time at night</li> <li>Child falls asleep within 20 minutes after</li> </ol> | going to bed | 3) Child falls asleep alone in own bed | 4) Child falls asleep in parent's or sibling's bed | 5) Child needs parent in the room to fall asleep | 6) Child struggles at bedtime (cries, refuses to | stay in bed, etc.) | <ol> <li>Child is afraid of sleeping in the dark</li> </ol> | 8) Child is afraid of sleeping alone | Child's usual amount of sleep each day (hours)<br>Child's usual amount of sleep each day | (minutes) | 9) Child sleeps too little | <br>Subcale 1: Bedtime Resistance | Subscale 2: Sleep Onset Delay | Subscale 8: Daytime Sleepiness | Total Sleep Disturbance Score |
| Category | Bedtime | | | | | | | | | | Sleep Behavior | | | Subscale and Total | Scores | | |
| Date of Assessment<br>(Study Day) | DDMMMYYYY (XX) | | | | | | | | | | | | | | | | |
| Study<br>Visit | XXXXXX | | | | | | | | | | | | | | | | |
| Treatment<br>[1] | XXXXXX XXXXXX XX-XXX | | | | | | | | | | | | | | | | |
| Subject<br>ID | XX-XX | | | | | | | | | | | | | | | | |

Note: Study day is calculated relative to the date of first dose of study drug. Assessments that are marked as Not Done are not included in the listing.

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

Programming Note: Continued for other categories and assessments. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment



Listing 16.2.7.1 Adverse Events All Subjects

| Severity/ Outcome/ Study Drug Action Taken/ Serious?// Abuse Other Action Taken Criteria Met Related? XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|
| Start Date (Study Day)/ End Date (Study Day)/ DDMMMYYYY/ DDMMMYYYYY/ Ongoing |
| System Organ Class/ Preferred Term/ Verbatim Term XXXXXXXXXXXXXXX XXXXXXXXXXXX XXXXXX |
| TEAE? |
| Subject ID Treatment TEAE? (1) (XX-XX XXXXXX XXX XXXXXXX XXX |
| Subject ID XXX-XX |

Abbreviation: TEAE = Treatment emergent adverse event.

Note: Study day is calculated relative to the date of first dose of study drug. AEs were coded using MedDRA version 19.1. A TEAE is any adverse event with an onset date/time between the initiation of study drug and 5 days after the last dose of study drug. This will include any AE with onset prior to initiation of study drug and increased severity after the treatment

1] Treatment is based on treatment received. The dose received at the beginning of the treatment-phase, or the last dose received if the subject discontinued from the study during the treatment-phase, is presented. \* = subject was down-titrated due to tolerability issues.

[2] Abuse-related AEs include the following MedDRA Preferred Terms: Euphoric mood; Elevated mood; Feeling abnormal; Feeling drunk; Feeling of relaxation; Dizziness; Thinking abnormal; Hallucination; Inappropriate affect; Somnolence; Mood disorders and disturbances; psychosis; aggression; confusion and disorientation; drug tolerance; habituation; drug folerance; withdrawal syndrome; substance-related disorders.

"Other" with the text. If Serious? is Yes, concatenate all serious criteria marked as Yes with a semicolon. If no events meet the criteria for display, present "No events are reported." Programming note: "Other Action Taken" will be either None, Medication Required, Relevant Procedure, or Other; if specify text is needed, concatenate "Relevant Procedure:" or SOC & PT text should be in proper case in table, as shown in the shell. Ensure correct MedDRA version is printed in footnote. Since treatment groups presented are based on the dose (mg) received at the beginning of the treatment-phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column.



Listing 16.2.8.1.1 Clinical Laboratory Data: Hematology All Subjects

| Comments/Reason<br>Not Done | × |
|---|---|
| Comments/<br>Not Done | XXXX |
| Accession<br>Number | ********** |
| Reference<br>Range Flag | × |
| Reference<br>Range [3] | \$\$\$\$\$\$\$\$\$<br>!!!!!!!!!!<br>********* |
| Change<br>from<br>Baseline [2] | **** |
| Standard<br>Results | ××××××× |
| Date of Assessment<br>(Study Day) | DDMMMYYYYY (X) |
| Study Visit | *********** |
| reatment [1] Parameter (unit) | Red Blood Cell Count |
| Treatment [1] | ××××××××××××××××××××××××××××××××××××××× |
| Subject<br>ID | ×××× |

Abbreviations: A = abnormal; CS = clinically significant; H = high; L = low; ND = not done.

Note: Study day is calculated relative to the date of first dose of study drug.

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment-Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

[2] Baseline is the Screening Visit 01A for new subjects and either the Screening Visit 01B or the last KP415.E01 Study Visit for roll-over subjects [3] Reference range is used to identify potentially clinically significant laboratory values.

Programming note: update abbreviations to reflect actual data. If test was not done, set results to ND; make sure last column is populated accordingly. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column.



Listing 16.2.8.1.2 Clinical Laboratory Data: Serum Chemistry All Subjects

(Same shell as Listing 16.2.8.1)

Listing 16.2.8.1.3 Clinical Laboratory Data: Urinalysis All Subjects

(Same shell as Listing 16.2.8.1; remove "(unit)" from 2nd column header)

Listing 16.2.8.1.4
Clinical Laboratory Data: Urine Drug Screen and Pregnancy Tests
All Subjects

(Same shell as Listing 16.2.8.1; remove "(unit)" from 2nd column header; do not display Reference Range or Accession number columns)



Listing 16.2.8.2 Vital Signs All Subjects

| | BMI | $(kg/m^2)$ | ×.× | | | | |
|---|---|---|---|---|---|---|---|
| BSA | $(m^2)$ | [2] | ××× | | | | |
| | Weight | (kg) | ×× | ×× | × | Q | × |
| | Height | (cm) | ××× | | | | |
| Sitting Blood | Pressure (mmHg) | Diastolic | × | × | × | Q | × |
| Sitting | | Systolic | × | × | × | Q | × |
| | Respiratory Rate | (breaths/min) | × | × | × | QN | × |
| | Pulse Rate | (beats/min) | × | × | × | Q | × |
| | Temp | (C) | ×× | ××× | ××× | 2 | XXX |
| Date of | Assessment | (Study Day) | _ | _ | _ | DDMMMYYYY (X) | DDMMMYYYY (X) |
| | Study | Visit | XXXXX | XXXXX | XXXXX | XXXXX | XXXXX |
| | Treatment | [1] | XXXXX | | | | |
| | Subject | D | XXXXX | | | | |

Abbreviation: BMI = Body Mass Index; BSA = body surface area; ND = not done.

Note: Study day is calculated relative to the date of first dose of study drug.

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

[2] BSA = $\sqrt{[\text{height(cm)} * \text{weight(kg)}]/3600}$ 

Programming Note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column.



Listing 16.2.8.3 12-Lead Electrocardiogram (ECG) Quantitative Results All Subjects

| Comments | | | | | | | | | XXXXXXXX |
|---|---|---|---|---|---|---|---|---|---|
| QTcF Interval<br>(msec) | × | ×× | × | × | × | ×× | | × | ××× |
| QT Interval<br>(msec) | × | ×× | × | × | × | × | | × | ××× |
| RR Interval (msec) | XX | XX | XX | X | × | XX | | × | ××× |
| Heart Rate<br>(bpm) | × | ×× | × | × | × | × | | × | ××× |
| Investigator<br>Interpretation | XXXXXXX | XXXXXXXXXX | XXXXXXXX | xxxxxxx | XXXXXXXXXX | XXXXXXXX | | XXXXXXX | XXXXXXXXXX |
| Date/Time of ECG<br>(Study Day) | DDMMMYYYY/ | DDMMMYYYY (X) | DDMMMYYYYY (X) | DDMMMYYYYY (X) | DDMMMYYYYY (X) | /AAAAAAAAAAAAAAAAAAAAAAAAAAAAAAAAAAAAA | (X)<br>QN<br>ND (X) | DDMMMYYYY/ | DDMMMYYYY/<br>hh:mm (X) |
| Study<br>Visit | XXXXX | XXXXX | XXXXX | XXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX | XXXXXX |
| Treatment [1] | XXXXXX | | | | | | | XXXXXX | |
| Subject ID | XXXXX | | | | | | | XXXXX | |

Abbreviation: HR = heart rate; ND = not done.

Note: Study day is calculated relative to the date of first dose of study drug.

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

Programming note: if assessment not done at a visit, put 'ND' in the date column. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column. Add columns for any additional parameters provided by the central reader.

AD-ST-33.05 Effective date: 22-Jan-2018

Version 0.1 | 07-Jun-2018 | AD-PR-109.01 Effective date: 26-Jun-2017




Listing 16.2.8.4 Columbia-Suicide Severity Rating Scale (C-SSRS) All Subjects

| Result | | XX |
|---|---|---|
| | * * * * | × × × × + × |
| Assessment | Wish to be dead If yes, describe: 2. Non-Specific Active Suicidal Thoughts If yes, describe: 3. Active Suicidal Ideation with Any Methods (not Plan) without Intent to Act If yes, describe: If yes, describe: Active Suicidal Ideation with | Some intent to Act, without Specific Plan If yes, describe: 5. Active Suicidal Ideation with Specific Plan and Intent If yes, describe: Was the answer to "1. Wish to be dead" and/or "2. Non-Specific Active Suicidal Thoughts" equal to "Yes"? Most Severe Ideation Type # (1-5) Description of Ideation |
| Category | Suicidal Ideation | Intensity of Ideation |
| Reference Period | Lifetime | |
| Date/Time<br>of Assessment<br>(Study Day) | DDMMMYYYY/<br>HH:MM (XX) | |
| Study Visit | × | |
| Treatment [1] | ××××× | |
| Subject<br>ID | ×××× | |

Note: Study day is calculated relative to the date of first dose of study drug. Assessments that are marked as Not Done are not included in the listing.
[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues. Programming Note: Continued for other categories and assessments. Screening and Baseline time points will have Lifetime and Past 6 months test periods. Other time points will have "Since last visit" test period. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column.


Listing 16.2.8.5 Physical Examination All Subjects

| Subject | | Study | Exam Date | | | | |
|---|---|---|---|---|---|---|---|
| | Treatment [1] | Visit | (Study Day) | Body System | Result | Abnormal Findings | Abnormal Findings Clinically Significant? |
| XXXXX | XX XXXXXXX XXX | XXXXXX | DDMMMYYYY | General | Normal | | |
| | | | (X-) | Appearance | | | |
| | | | | Skin | Abnormal | XXXXXXX | No |
| | | | | Head and Neck | Normal | | |
| | | | | Lymph Nodes | Normal | | |
| | | | | Thyroid | Normal | | |
| | | | | Musculoskeletal | Normal | | |
| | | | | Extremeties | Normal | | |
| | | | | Cardiovascular | Normal | | |
| | | | | Lungs | Normal | | |
| | | | | Abdomen | Normal | | |
| | | | | Neurological | Normal | | |

Note: Study day is calculated relative to the date of first dose of study drug.
[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

Programming note: Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the to data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column.



Listing 16.2.8.6 Prior and Concomitant Medications All Subjects

| Route/<br>Frequency | /XXXXXXXX | <b>***</b> | | | | |
|---|---|---|---|---|---|---|
| Route/<br>Freque | × | { | | | | |
| Dose (unit) /<br>Total Daily Dose | /(xxx) xxx | <b>*</b> | / (xxx) xxx | *** | / (xxx) xxx | *** |
| Start Date (Study Day)/<br>End Date (Study Day) | DDMMMYYYY (X)/ | DDMMMYYYY (X) | DDMMMYYYY (X)/ | Ongoing | DDMMMYYYY (X)/ | DDMMMYYYY (X) |
| ATC Class (Level 4)/<br>Preferred Term (ATC Level 5)/<br>Verbatim Term | /xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | \xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | /XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | /XXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| Reason for<br>Use | XXXXXXXX | | XXXXXXX | | XXXXXX | |
| Prior/<br>Concomitant Reason for<br>[2] Use | Prior | | Both | | Concomitant XXXX | |
| Subject ID Treatment [1] | XXXXXX | | | | | |
| Subject ID | XXXXXX XXXXXX | | | | | |

Abbreviation: ATC = anatomic therapeutic chemical; NA = Not applicable.

Note: Study day is calculated relative to the date of first dose of study drug. Medications were coded using WHO-DDE version September 2017.
[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

[2] Prior indicates medication that was started and stopped prior to dosing of study drug. Concomitant indicates medication that started during the treatment period. Both indicates medication that was started prior to dosing of study drug and continued during the treatment period. Programming note: If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX" but just "XXXXXXX"). Sort by subject, start date/time, end date/time, ATC level 4 & PT. ATC & PT text should be in proper case in table, as shown in the shell. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the

treatment in the treatment column.



Listing 16.2.8.7 Lifetime History of ADHD Treatment All Subjects

| End Date<br>(Study Day) | XXXXXXXX<br>(XXX) | XXXXXXXX<br>(XXX) | XXXXXXXX<br>(XXX) |
|---|---|---|---|
| Ongoing? | × | × | × |
| Was this<br>Medication<br>Started<br>Within the<br>Last 14<br>Days? | ×× | ×× | ×× |
| Start Date<br>(Study Day) | XXXXXXXX<br>(XXX) | XXXXXXX<br>(XXX) | XXXXXXX<br>(XXX) |
| Reason for<br>Use | XXXXXXX XXXXXXX | XXXXXX | XXXXXX |
| Frequency | XXXXXXX | XXXXXX | XXXXXX |
| Route | XXXXXX | XXXXXX | XXXXXX |
| Dose<br>(Dose<br>Unit) | XXXXX) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXX) |
| ADHD Drug<br>Class | XXXXXX | XXXXXX | XXXXXX |
| Subject Treatment Medication/Therapy ADHD Drug<br>ID [1] Name Class | XXXXXXX XXXXXXX XXXXXXXX | XXXXXXX | ×××××× |
| Treatment<br>[1] | XXXXX | | |
| Subject<br>ID | XXXXX | | |

Abbreviation: ADHD = attention-deficit hyperactivity disorder; NA = Not applicable.

Note: Study day is calculated relative to the date of first dose of study drug.
[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

Programming note: If Dose unit, Route or Frequency is Other, display other specify text only (ie, do not display "Other: XXXXXX" but just "XXXXXX"). Sort by subject, start dater/time, end date/time, ADHD Drug Class, Medication/Therapy Name. ADHD Drug Class and Medication/Therapy Name text should be in proper case in table, as shown in the shell. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a

lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column.

Version 0.1 | 07-Jun-2018 | AD-PR-109.01 Effective date: 26-Jun-2017

AD-ST-33.05 Effective date: 22-Jan-2018



Listing 16.2.8.8 ADHD Medication Washout All Subjects

Abbreviations: ADHD = attention-deficit hyperactivity disorder.

[1] Treatment is based on treatment received. The dose received at the beginning of the Treatment Phase, or the last dose received if the subject discontinued from the study during the Treatment Phase, is presented. \* = subject was down-titrated due to tolerability issues.

Programming note: Sort by subject, start date, end date. Since treatment groups presented are based on the dose (mg) received at the beginning of the Treatment Phase, actual doses need to be determined from the data. If a subject receives a lower dose than planned due to tolerability, place an asterisk next to the treatment in the treatment column. If the subject was not reminded of the washout, concatenate reason like: "No: XXXXXXX".



**premier** research



Not Applicable



## **Appendix 1: Premier Research Library of Abbreviations**

| Abbreviation | Definition |
|--------------|---------------------------------------------------------|
| aCRF | annotated case report form |
| AD | associated documents |
| ADHD | attention-deficit hyperactivity disorder |
| ADHD-RS-5 | Attention-Deficit Hyperactivity Disorder Rating Scale 5 |
| ADR | adverse drug reactions |
| AE | adverse event |
| AESI | adverse events special interest |
| AIC | Akaike information criterion |
| ALT | alanine aminotransferase |
| ANCOVA | analysis of covariance |
| AR(1) | Autoregressive |
| AST | aspartate aminotransferase |
| ATC | anatomical therapeutic chemical |
| BLQ | beneath limit of quantification |
| BMI | body mass index |
| BSA | body surface area |
| CCGs | CRF completion guidelines |
| CD | compact disc |
| CDISC | clinical data interchange standards consortium |



| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| CEC | central ethics committee |
| CFR | code of federal regulations |
| CGI-I | Clinical Global Impressions–Improvement |
| CGI-S | Clinical Global Impressions–Severity |
| CI | confidence intervals |
| CIOMS | council for international organizations of medical sciences |
| CIP | clinical investigational plan |
| CM | clinical manager or centimeter |
| CMP | clinical monitoring plan |
| COV | close out visit |
| CRA | clinical research associate |
| CRF | case report form |
| CRO | contract research organization |
| CS | clinically significant or compound symmetry |
| CSHQ | Children's Sleep Habits Questionnaire |
| CSM | clinical supply manager |
| CSR | clinical study report |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CTA | clinical trial administrator |
| CTM | clinical trial manager |
| CTMS | clinical trial management system |



| Abbreviation | Definition |
|--------------|-------------------------------------------|
| DB | database |
| DBL | database lock |
| DBP | diastolic blood pressure |
| DCRF | data change request form |
| DDE | drug dispensing error form |
| DEA | drug enforcement administration |
| DIA | drug information association |
| DIS | data integration specification |
| DLT | dose limiting toxicity |
| DM | data management |
| DMB | data monitoring board |
| DMC | data monitoring committee |
| DML | data management lead |
| DMP | data management plan |
| DNA | deoxyribonucleic acid |
| DOB | date of birth |
| DS | document specialist |
| DSG | drug safety group |
| DSM | drug supply management (drug distributor) |
| DSMB | data safety monitoring board |
| DSP | data safety plan |



| Abbreviation | Definition |
|--------------|------------------------------------------|
| DSUR | development safety update report |
| DTS | data transfer specification |
| DVD | digital video disk |
| EC | ethics committee |
| ECD | edit check and derivation specifications |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EDC | electronic data capture |
| EMA | European medicines agency |
| EOS | end of study |
| ЕОТ | end of treatment |
| ET | early termination |
| eTMF | electronic trial master file |
| EU | European Union |
| FA | full analysis |
| FDA | food and drug administration |
| FMP | file management plan |
| FPFV | first patient first visit |
| FPI | first patient in |
| GCP | good clinical practice |
| GMP | good manufacturing practices |



| Abbreviation | Definition |
|--------------|------------------------------------------------|
| GPV | global pharmacovigilance |
| HEENT | Head, neck, eyes, ears, nose, mouth, and thoat |
| HR | heart rate |
| IB | investigator's brochure |
| IC or ICF | informed consent or informed consent form |
| ICH | international council for harmonization |
| ID | identification |
| IDM | independent drug monitoring |
| IEC | independent ethics committee |
| IM | investigator meeting |
| IMV | interim monitoring visit |
| IND | investigational new drug |
| INDSR | investigational new drug safety reports |
| IP | investigational product |
| IRB | institutional review board |
| IRF | inventory release file |
| IRR | infusion related reactions |
| IRT | interactive response technology |
| ISF | investigator site file |
| ITT | intent-to-treat |
| IVRS | interactive voice response system |



| Abbreviation | Definition |
|---|---|
| IWRS | interactive web response system |
| IxRS | interactive voice/web response system |
| kg | kilogram |
| KPI | key performance indicator |
| LAN | local area network |
| LDM | lead data manager |
| LMS | learning management system |
| LLOQ | lower limit of quantification |
| LOCF | last observation carried forward |
| LPI | last patient in |
| LPLV | last patient last visit |
| LPO | last patient out |
| LS | least squares |
| MAAP | medical affairs and pharmacovigilance teams |
| MAH | marketing authorization holder |
| MedDRA | medical dictionary for regulatory activities |
| mg | milligram |
| MHRA | medicines and healthcare products regulatory agency |
| MINI-KID | Mini International Neuropsychiatric Interview for Children and Adolescents |
| mL | milliliter |



| Abbreviation | Definition |
|--------------|---------------------------------------|
| MM | medical monitor |
| MMP | medical monitoring plan |
| MMRM | mixed effect model repeat measurement |
| МРН | methylphenidate |
| MTD | maximum tolerated dose |
| MVR | monitoring visit report |
| N | number |
| NA | not applicable |
| NCS | non-clinically significant |
| NF | non-functional |
| PD | protocol deviation |
| PDGP | protocol deviation guidance plan |
| PE | physical examination |
| pH | hotential hydrogen |
| PI | principal investigator |
| PIN | personal identification number |
| PK | pharmacokinetic |
| PKAP | pharmacokinetic analysis plan |
| PM | project manager |
| PMP | project management plan |
| PP | per-protocol |



| Abbreviation | Definition |
|---|---|
| PRIMS | Premier Research information management system |
| PS | project specialist |
| PT | preferred term or Prothrombin Time |
| PTT | Prothrombin Thromboplastin Time |
| PV | pharmacovigilance |
| PVG | pharmacovigilance group |
| QA | quality assurance |
| QARC | quality assurance, risk and compliance |
| QC | quality control |
| QOL | quality of life |
| QTcF | Time between the start of the Q wave and the end of the T wave (QT interval) in the heart's electrical cycle, corrected for heart rate with Fridericia's formula |
| ROT | record of training |
| RR | respiratory rate or relative rate |
| RSM | regional site monitor |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS® | a software system used for data analysis |
| SBP | systolic blood pressure |
| SC | study coordinator |
| SCR | software change request |



| Abbreviation | Definition |
|--------------|--------------------------------------------------------|
| SD | standard deviation |
| SDS | study design specifications |
| SDTM | study data tabulation model |
| SDV | source data verification |
| SECC | self-evident correction conventions |
| SECP | self-evident correction plan |
| SF | screen failure |
| SFT or SFTP | secure file transfer or secure file transfer plan |
| SIV | site initiation visit |
| SLA | service level agreement |
| SMP | safety management plan |
| SOC | system organ class |
| SOP | standard operating procedure |
| SOW | statement of work |
| SQV | site qualification visit |
| SUA | start-up associate |
| SUSAR | suspected, unexpected, serious adverse (drug) reaction |
| TA | trial assistant |
| TEAE | treatment-emergent adverse event |
| TMF | trial master file |
| TOM | task ownership matrix |





| Abbreviation | Definition |
|--------------|----------------------------------------------------|
| TSH | thyroid stimulating hormone |
| UAT | user acceptance testing |
| USA | United States of America |
| UTC | universal coordinated time |
| VC | variance components |
| WAN | wide area network |
| WAR | work at risk |
| WG | working guideline |
| WHO | world health organization |
| WHO-DD | world health organization drug dictionary |
| WHO-DDE | world health organization drug dictionary enhanced |